CLINICAL TRIAL: NCT00814320
Title: Efficacy, Tolerability and Pharmacokinetic Comparison of Immune Globulin Intravenous (Human), 10% (GAMMAGARD LIQUID/KIOVIG) Administered Intravenously or Subcutaneously Following Administration of Recombinant Human Hyaluronidase (rHuPH20) in Subjects With Primary Immunodeficiency Diseases
Brief Title: Gammagard Liquid and rHuPH20 in PID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160603
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Efficacy and tolerability of subcutaneous (SC) infusions of immune globulin intravenous (IGIV), 10% with hyaluronidase (rHuPH20) after ramp-up
  Interventions: Biological: Recombinant human hyaluronidase (rHuPH20)+ immune globulin intravenous (IGIV)
- 2 (Experimental): Pharmacokinetics of intravenous (IV) infusions of immune globulin intravenous (IGIV), 10% and efficacy and tolerability of subcutaneous (SC) infusions of immune globulin intravenous (IGIV), 10% with hyaluronidase (rHuPH20) after ramp-up
  Interventions: Biological: Recombinant human hyaluronidase (rHuPH20)+ immune globulin intravenous (IGIV)

INTERVENTIONS:
Biological: Recombinant human hyaluronidase (rHuPH20)+ immune globulin intravenous (IGIV) — Comprises subjects previously participating in Study 160601, who now only complete Study Epoch 2 (subcutaneous [SC] infusions) as bioavailability/exposure for intravenous (IV) treatment was already obtained in Study 160601.
  Study Epoch 2: Dose (calculated) of rHuPH20 followed by dose (calculated) of IGIV, 10% by SC infusion. Treatment intervals and doses are to be increased as defined, until treatment interval is the same as the pre-study treatment interval for IV treatment (ramp-up).
  Other Names: HYQVIA
  Arms: 1
Biological: Recombinant human hyaluronidase (rHuPH20)+ immune globulin intravenous (IGIV) — Comprises all other subjects.
  Study Epoch 1: IV infusion of IGIV, 10% (same dose and frequency as pre-study) to determine pharmacokinetics.
  Study Epoch 2: Dose (calculated) of rHuPH20 followed by dose (calculated) of IGIV, 10% by SC infusion. Treatment intervals and doses are to be increased as defined, until treatment interval is the same as the pre-study treatment interval for IV treatment (ramp-up).
  Arms: 2

SUMMARY:
The purpose of the study is to develop a subcutaneous treatment option for participants with Primary Immunodeficiency Diseases (PID) that allows an administration of Immune Globulin Intravenous (Human), 10% at the same frequency as IV administration.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 2 years or older at the time of screening
* Written informed consent obtained from either the participant or the participant's legally acceptable representative prior to any study-related procedures and study product administration
* Participant has been diagnosed with a PID disorder requiring antibody replacement as defined by WHO criteria
* Participant has completed or is about to complete Baxter Clinical Study Protocol No. 160601 or has been receiving a regular IGIV-treatment at mean intervals of 21 ± 3 days or 28 ± 3 days, or SC at mean intervals of 5 to 16 days, over a period of at least 3 months prior to enrollment at a minimum dose of 300 mg/kg BW/4 weeks
* Participant has a serum trough level of IgG > 4.5 g/L at the last documented determination
* If female of childbearing potential, participant presents with a negative urine pregnancy test and agrees to employ adequate birth control measures for the duration of the study
* Participant is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Participant has a known history of or is positive at enrollment or screening for one or more of the following: Hepatitis B surface antigen (HbsAg), polymerase chain reaction (PCR) for Hepatitis C Virus (HCV), PCR for Human immunodeficiency virus (HIV) Type 1/2
* Participant has levels of alanine aminotransferase (ALT) or aspartate amino transferase (AST) > 2.5 times the upper limit of normal for the testing laboratory
* Participant has persistent severe neutropenia (defined as an absolute neutrophil count [ANC] <= 500/mm3)
* Participant has creatinine clearance (CLcr) values, calculated according to the formula below, which are < 60% of normal for age and gender for males: CLcr = [(140 - Age(years)) * (body weight (kg))] / [72 * (serum creatinine (mg/dL))] for females: CLcr = [(140 - Age(years)) * (body weight(kg)) * 0.85] / [72 * (serum creatinine (mg/dL))]
* Participant has been diagnosed with, or has a malignancy (other than adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) within the last 12 months prior to enrollment; participants treated with immunosuppressive chemotherapeutic agents during this period are excluded
* Participant has a history of thrombotic episodes (including deep vein thrombosis, myocardial infarction, cerebrovascular accident, pulmonary embolism) within the last 12 months
* Participant has abnormal protein loss (protein losing enteropathy, nephrotic syndrome)
* Participant has anemia that would preclude phlebotomy for laboratory studies
* Participant has received any blood or blood product other than an IGIV, SC immunoglobulin, immune serum globulin (ISG) preparation, or albumin within the 6 months prior to enrollment
* Participant has an ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following IGIV, SC immunoglobulin, and/or ISG infusions
* Participant has immunoglobulin A (IgA) deficiency and known anti IgA antibodies
* Participant is on preventative (prophylactic) antibiotics and cannot stop antibiotics at the time of enrollment
* Participant has active infection who started on antibiotic therapy for the treatment of infection within 7 days prior to screening
* Participant has a bleeding disorder or is on anti-coagulation therapy that results in a platelet count less than 20,000/μL or International Normalized Ration (INR) > 2X control, or who, in the opinion of the investigator would be at significant risk of increased bleeding or bruising as a result of SC therapy
* Participant has total protein > 9 g/dL and participants with myeloma, macroglobulinemia (IgM) and paraproteinemia
* Participant has a known allergy to hyaluronidase
* If female, participant is pregnant or lactating at the time of study enrollment
* Participant has participated in another clinical study involving an investigational product (IP) or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an IP or device during the course of this study; exception: Baxter Study No. 160601
* Severe dermatitis that would preclude adequate sites for safe product administration

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-12-18 (Actual); Primary Completion 2010-11-11 (Actual); Study Completion 2010-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (14):
- United States (13):
  - Cypress, California
  - Irvine, California
  - Los Angeles, California
  - San Francisco, California
  - Centennial, Colorado
  - North Palm Beach, Florida
  - Atlanta, Georgia
  - Hinsdale, Illinois
  - Omaha, Nebraska
  - The Bronx, New York
  - Dallas, Texas
  - Galveston, Texas
  - Milwaukee, Wisconsin
- Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Wasserman RL, Melamed I, Stein MR, Engl W, Sharkhawy M, Leibl H, Puck J, Rubinstein A, Kobrynski L, Gupta S, Grant AJ, Ratnayake A, Richmond WG, Church J, Yel L, Gelmont D. Long-Term Tolerability, Safety, and Efficacy of Recombinant Human Hyaluronidase-Facilitated Subcutaneous Infusion of Human Immunoglobulin for Primary Immunodeficiency. J Clin Immunol. 2016 Aug;36(6):571-82. doi: 10.1007/s10875-016-0298-x. Epub 2016 May 25. PMID 27220317
- [Result] Wasserman RL, Melamed I, Stein MR, Gupta S, Puck J, Engl W, Leibl H, McCoy B, Empson VG, Gelmont D, Schiff RI; IGSC, 10% with rHuPH20 Study Group. Recombinant human hyaluronidase-facilitated subcutaneous infusion of human immunoglobulins for primary immunodeficiency. J Allergy Clin Immunol. 2012 Oct;130(4):951-7.e11. doi: 10.1016/j.jaci.2012.06.021. Epub 2012 Jul 28. PMID 22846381
- [Derived] Wasserman RL, Gupta S, Stein M, Rabbat CJ, Engl W, Leibl H, Yel L. Infection rates and tolerability of three different immunoglobulin administration modalities in patients with primary immunodeficiency diseases. Immunotherapy. 2022 Mar;14(4):215-224. doi: 10.2217/imt-2021-0256. Epub 2021 Dec 21. PMID 34931880

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted 14 clinical sites in the United States and 1 clinical site in Canada.
Pre-assignment Details: 89 participants who enrolled were screened. Of these, 2 withdrew before treatment (both were screen failures)
Groups:
- 2 to <12 Years: The same as the other study arm/group (please see "12 Years and Older", due to character limitation) with the exception of the pharmacokinetic assessment that was done. For participants aged 2 to <12 years, immunoglobulin G (IgG) trough levels only were assessed in order to avoid multiple blood drawings in small children.
- 12 Years and Older: EPOCH 1: Pharmacokinetics (PK) of intravenous (IV) administration of immune globulin intravenous (IGIV), 10%. Participants who previously participated in Study 160601 entered this study directly to Epoch 2 ramp-up. PK data collected during IV treatment in Study 160601 was compared with PK data from subcutaneous (SC) treatment during this study. EPOCH 2 RAMP-UP ("ramp-up"):Treatment intervals/ doses used for initial SC infusions of IGIV, 10% were slowly increased during first weeks of treatment to allow participants to adjust to increasing volume administered SC. Prior to SC infusions, recombinant human hyaluronidase (rHuPH20) was administered at a minimum dose of 75 U/g IgG. EPOCH 2 after RAMP-UP: Participants were treated SC with IGIV, 10% with rHuPH20 at 108% of IV dose from Epoch 1 (or from study 160601). Prior to SC infusions, rHuPH20 was administered at a minimum dose of 75 U/g IgG. Aim was to treat participants SC at same intervals (ie, every 3 or 4 weeks) as treated IV.
Period: Epoch 1 (IV Treatment)
Arm/Group | 2 to <12 Years | 12 Years and Older
Started | 14 | 73
Completed | 13 | 71
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Participant missed 2 consecutive doses | 0 | 2
Period: Between Epoch 1 (IV) and Epoch 2 Ramp-up
Arm/Group | 2 to <12 Years | 12 Years and Older
Started | 13 | 71
Completed | 13 | 70
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Epoch 2 Ramp-up ("Ramp-up")
Arm/Group | 2 to <12 Years | 12 Years and Older
Started | 13 | 70
Completed | 11 | 70
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Geographic Factor | 1 | 0
Period: Epoch 2 After Ramp-up (SC/rHuPH20)
Arm/Group | 2 to <12 Years | 12 Years and Older
Started | 11 | 70
Completed | 8 | 60 (Three participants who switched to safety follow-up remained in the study.)
Not Completed | 3 | 10
Not completed — Adverse Event | 1 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Subject Felt Increased Infections on SC | 0 | 1
Not completed — Switched to safety follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- 12 Years and Older: EPOCH 1: Pharmacokinetics (PK) of Intravenous (IV) treatment and efficacy and tolerability of Subcutaneous (SC) infusions Recombinant human hyaluronidase (rHuPH20) + immune globulin intravenous (IGIV). Participants who previously participated in Study 160601 entered this study at Epoch 2. PK data collected during IV treatment in Study 160601 were used for comparison with PK data from SC treatment during this study (160603). EPOCH 2: (ramp-up and After ramp-up). Participants were treated SC with GAMMAGARD LIQUID/KIOVIG at 108% of IV dose from Epoch 1 or Study 160601. 108% was derived from PK data from Study 160602. Prior to SC infusions, rHuPH20 was administered at a minimum dose of 75 U/g IgG. Treatment intervals and doses used for initial infusions were gradually increased during first weeks of treatment (ramp-up), to allow participants to adjust to increasing volume administered SC. Aim was to treat participants SC at same intervals (ie, every 3 or 4 weeks) as treated IV.
- Total: Total of all reporting groups
Arm/Group | 2 to <12 Years | 12 Years and Older | Total
Number analyzed (Participants) | 14 | 73 | 87
Age, Continuous [Median (Full Range); unit: years] | 8.0 [4 to 11] | 44.0 [12 to 78] | 35.0 [4 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 37 | 43
  Male | 8 | 36 | 44
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 72 | 86
  Canada | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Validated Acute Serious Bacterial Infection (VASBI) Rate
Description: Serious acute bacterial infections include bacteremia/sepsis, bacterial meningitis, osteomyelitis/septic arthritis, bacterial pneumonia, and visceral abscess that are caused by a recognized bacterial pathogen. VASBI rate is the mean number of VASBIs per participant per year, recorded for SC Administration of IGIV, 10%, with rHuPH20 after ramp-up, only. The mean number of VASBIs per participant per year and the 99% upper confidence limit for the acute serious bacterial infection rate were calculated using a Poisson model to account for the length of the observation periods per participant.
Time Frame: Throughout the study period (17 months)
Measure: Number; unit: Estimated infections/year
Groups:
- Full Analysis Data Set (FADS): All participants who had been exposed to either or both study drugs and who provided data for the primary endpoint for any period of time.
Arm/Group | Full Analysis Data Set (FADS)
Number analyzed (Participants) | 81
Estimated infections/year | 0.025
Statistical Analysis 1: Comparison: Full Analysis Data Set (FADS); For SC Administration of IGIV, 10%, with rHuPH20 after ramp-up, only; Test type: Superiority or Other; p < 0.0001, Poisson — Testing the null hypothesis of 1 VASBI/year against a one-sided alternative at the 0.01 level of statistical significance; Poisson = 0.025, 99% CI 1-sided [upper limit 0.046]

2. Secondary Outcome: Bioavailability (AUC) of IgG After Administration of IGIV, 10% Given Via IV or SC With rHuPH20 in Participants ≥12 Years
Description: Bioavailability expressed as pharmacokinetic (PK) equivalence of immunoglobulin (IgG) in terms of ratio of Area Under the Concentration Curve (AUC)/Week after administration of immune globulin intravenous (IGIV), 10% given via subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up to intravenous (IV) route, i.e. ratio of AUC/week of SC/rHuPH20 versus IV administration of IGIV, 10%. Expressed as a percentage.
Time Frame: PK AUC evaluations: (IV: before infusion #4 [for 3-week treatment interval] or infusion #3 [for 4-week treatment interval];SC: before last SC infusion) 60 minutes pre-infusion up to 28 days (+/-2 days) post-infusion
Population: Participants ≥ 12 years exposed to either or both study drugs with AUC measurements at the following time points: Pre-infusion and 30-minutes post-infusion (Day 0) IV- Days 1, 4, 9, 14, 21, 28* SC- Days 1, 3, 5, 9, 14, 21, 28* *Measurements at Day 28 for the 4-week treatment interval only
Measure: Number (90% Confidence Interval); unit: Percentage
Groups:
- % Ratio IgG AUC/Week of SC/ IV: Percentage Ratio of IgG AUC (/Week) after SC administration with rHuPH20/ IgG AUC (/Week) after IV administration of IGIV, 10%
Arm/Group | % Ratio IgG AUC/Week of SC/ IV
Number analyzed (Participants) | 58
Percentage | 93.3 [91.4 to 95.2]

3. Secondary Outcome: Bioavailability (Trough Levels) of IgG After Administration of IGIV, 10% Given Via IV or SC With rHuPH20 in Participants Aged 2 to < 12 Years
Description: Bioavailability expressed as pharmacokinetic (PK) equivalence of immunoglobulin (IgG) in terms of trough levels after administration of immune globulin intravenous (IGIV), 10% given via subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up to intravenous (IV) route, i.e. ratio of AUC/week of SC/rHuPH20 versus IV administration of IGIV, 10%. Expressed as a percentage.
Time Frame: IgG trough levels measured at baseline and on day of each 3- or 4-week infusion for infusion for IV and SC (except during ramp-up for SC) and at end of study visit
Population: Participants aged 2 to < 12 years exposed to either or both study drugs with available IgG trough level measurements
Measure: Number (95% Confidence Interval); unit: Percentage
Groups:
- %Ratio IgG Trough Level of SC/IV: Percentage Ratio IgGTrough Level after SC administration with rHuPH20/IgG versus after IV administration of IGIV, 10% for participants aged 2 to < 12 years
Arm/Group | %Ratio IgG Trough Level of SC/IV
Number analyzed (Participants) | 11
Percentage | 103.8 [97.5 to 115.4]

4. Secondary Outcome: Bioavailability (AUC) of IgG After SC Administration of IGIV, 10%, Given With and Without rHuPH20
Description: Bioavailability of immunoglobulin (IgG) after subcutaneous (SC) administration of immune globulin intravenous (IGIV), 10%, with and without recombinant human hyaluronidase (rHuPH20) (from current study 160603 and study 160601, respectively), as measured by ratio of AUC of IgG per dose/kg with versus without rHuPH20. Expressed as a percentage. This was analysed for participants in Stratum A , participants in Stratum B and for all participants who received IGIV, 10% via SC administration (Stratum A plus Stratum B): Stratum A: Participants who provided data both on SC with AND without rHuPH20 ie, participants who participated in both studies 160601 and 160603; Stratum B: Participants who provided data on SC with OR without rHuPH20, but not on both (participants who participated in study 160601 OR 160603, but not in both studies).
Time Frame: PK: 160603 (IV: before infusion (inf.) #4 [3-week treatment interval] or inf. #3 [4-week treatment interval];SC: before last SC inf.) 1 hour pre-inf. ≤28 days (+/-2 days) post-inf.; 160601- 1 hour pre-inf. (before inf. #8) ≤7 days (+/-1 day) post-inf.
Population: Participants in the Full Analysis Data Set aged ≥ 12 years from the current study (160603) and prior Baxter study 160601 who received IGIV, 10% via SC administration
Measure: Number (90% Confidence Interval); unit: Percentage
Groups:
- Ratio IgG AUC of SC With and Without rHuPH20: Percentage Ratio of IgG AUC (dose per kg) with and without rHuPH20 for SC administration of IGIV, 10%
Arm/Group | Ratio IgG AUC of SC With and Without rHuPH20
Number analyzed (Participants) | 73
Percentage
  Participants in Stratum A (N=19) | 118.7 [113.6 to 124.1]
  Participants in Stratum B (N=54) | 133.6 [118.3 to 150.8]
  Total Participants (N=73) | 120.4 [115.5 to 125.5]

5. Secondary Outcome: Annual Rate of All Infections Per Participant
Description: Annual rate of all infections per participant after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up. Point estimates and 95% CIs for the annual rates will be calculated using a Poisson model and the same methodology including allowance for over-dispersion as described for the primary endpoint.
Time Frame: Throughout the study period (17 months)
Population: Full Analysis Data Set
Measure: Number (95% Confidence Interval); unit: Estimated infections/year
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10%, With rHuPH20 After Ramp-up
Number analyzed (Participants) | 81 | 81
Estimated infections/year | 4.51 [3.50 to 5.69] | 2.97 [2.51 to 3.47]

6. Secondary Outcome: Trough Levels of IgG After Administration of IGIV, 10% Given Via IV or SC With rHuPH20
Description: Trough levels of immunoglobulin (IgG) after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up
Time Frame: IgG trough levels measured at baseline and on day of each 3- or 4-week infusion for IV and SC (except during ramp up for SC) and at end of study visit.
Population: Full Analysis Data Set
Measure: Median (95% Confidence Interval); unit: g/L
Arm/Group | Participants Aged 2 to <12 Years | Participants ≥12 Years
Number analyzed (Participants) | 11 | 70
g/L
  end of IV part | 9.63 [8.29 to 13.60] | 10.40 [9.63 to 11.4]
  end of SC with rHuPH20 part | 9.95 [7.87 to 15.00] | 10.70 [9.46 to 11.80]

7. Secondary Outcome: Trough Levels of IgG Subclasses After Administration of IGIV, 10% Given Via IV or SC With rHuPH20
Description: Trough levels of immunoglobulin (IgG) subclasses after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up by IgG subclasses 1 to 4 at end of IV treatment and end of SC treatment with rHuPH20 IgG subclass 1 (IgG 1) IgG subclass 2 (IgG 2) IgG subclass 3 (IgG 3) IgG subclass 4 (IgG 4)
Time Frame: IgG subclasses (1-4) trough levels measured at baseline and on day of each 3- or 4-week infusion for infusion for IV and SC (except during ramp up for SC) and at end of study visit
Population: Participants who have been exposed to either or both study drugs with available IgG subclass trough level measurements
Measure: Median (95% Confidence Interval); unit: mg/dL
Arm/Group | Participants Aged 2 to <12 Years | Participants ≥ 12 Years
Number analyzed (Participants) | 11 | 70
mg/dL
  IgG 1 end of IV treatment (N=11,69) | 490.0 [414.0 to 752.0] | 574.0 [514.0 to 638.0]
  IgG 1 end of SC/rHuPH20 treatment (N=11,70) | 455.0 [411.0 to 805.0] | 548.0 [513.0 to 602.0]
  IgG 2 end of IV treatment (N=11,69) | 327.0 [250.0 to 538.0] | 360.0 [334.0 to 390.0]
  IgG 2 end of SC/rHuPH20 treatment (N=11,70) | 315.0 [280.0 to 550.0] | 339.0 [318.0 to 374.0]
  IgG 3 end of IV treatment (N=11,69) | 35.0 [27.0 to 66.0] | 32.0 [27.0 to 37.0]
  IgG 3 end of SC/rHuPH20 treatment (N=11,70) | 49.0 [26.0 to 83.0] | 36.0 [32.0 to 43.0]
  IgG 4 end of IV treatment (N=11,69) | 24.0 [16.0 to 55.0] | 14.0 [13.0 to 20.0]
  IgG 4 end of SC/rHuPH20 treatment (N=11,70) | 23.0 [15.0 to 57.0] | 15.0 [13.0 to 19.0]

8. Secondary Outcome: Antibody Levels to Tetanus (Clostridium Tetani Toxoid)
Description: Antibody levels to Tetanus (Clostridium tetani toxoid) after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) at end of IV treatment and end of SC treatment with rHuPH20
Time Frame: IV: At baseline; SC/rHuPH20: at baseline then at infusion #1 at ramp-up and at infusions #5, 9, 13 (for 3-week treatment interval) and infusions #4, 7, 10 (for 4-week treatment interval), SC: end of SC treatment and at end of study visit
Population: Participants in Full Analysis Data Set with available specific antibody test results
Measure: Median (95% Confidence Interval); unit: IU/mL
Arm/Group | Participants Aged 2 to <12 Years | Participants ≥ 12 Years
Number analyzed (Participants) | 10 | 70
IU/mL
  End of IV treatment (N=7,25) | 2.230 [0.0640 to 4.230] | 2.320 [1.810 to 2.710]
  End of SC/rHuPH20 treatment (N=10,70) | 2.580 [0.990 to 3.810] | 2.525 [2.270 to 2.850]

9. Secondary Outcome: Antibody Levels to Haemophilus Influenzae
Description: Antibody levels to Haemophilus influenzae after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) at end of IV treatment and end of SC treatment with rHuPH20
Time Frame: as for outcome 8
Population: Participants in Full Analysis Data Set with available specific antibody test results
Measure: Median (95% Confidence Interval); unit: μg/mL
Arm/Group | Participants Aged 2 to <12 Years | Participants ≥ 12 Years
Number analyzed (Participants) | 10 | 70
μg/mL
  Influenza antibody end of IV treatment (N=7,24) | 2.11 [1.59 to 13.52] | 2.36 [2.05 to 3.05]
  Influenza antibody end of SC treatment (N=10,70) | 1.97 [1.69 to 4.94] | 2.58 [2.30 to 2.95]

10. Secondary Outcome: Antibody Levels to Measles
Description: Antibody levels to measles after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) at end of IV treatment and end of SC treatment with rHuPH20
Time Frame: as for outcome 8
Population: Participants in the Full Analysis Data Set with available specific antibody test results
Measure: Median (95% Confidence Interval); unit: Titer
Arm/Group | Participants Aged 2 to <12 Years | Participants ≥ 12 Years
Number analyzed (Participants) | 10 | 70
Titer
  Measles antibody end of IV treatment (N=0,1) | NA [NA to NA] — No entry in this category/arm | 64.0 [NA to NA] — One entry in this category/arm
  Measles antibody end of SC treatment (N=10,70) | 768.0 [256.0 to 2048.0] | 1024.0 [512.0 to 1024.0]

11. Secondary Outcome: Antibody Levels to Hepatitis B
Description: Antibody levels to hepatitis B after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) with recombinant human hyaluronidase (rHuPH20) at end of IV treatment and end of SC treatment with rHuPH20
Time Frame: as for outcome 8
Population: Participants in the Full Analysis Data Set with available specific antibody test results
Measure: Median (95% Confidence Interval); unit: mIU/mL
Arm/Group | Participants Aged 2 to <12 Years | Participants ≥ 12 Years
Number analyzed (Participants) | 10 | 70
mIU/mL
  Hepatitis B antibody end IV treatment (N=6,25) | 212.9 [59.5 to 291.5] | 222.8 [190.3 to 289.4]
  Hepatitis B antibody end of SC treatment (N=10,70) | 242.2 [125.5 to 871.9] | 249.2 [225.0 to 289.3]

12. Secondary Outcome: IgG Minimum Plasma Concentration (C_min) for Participants Aged 12 Years and Older
Description: Minimal immunoglobulin (IgG) concentration after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and Older
Time Frame: PK evaluations: (IV: before infusion #4 [for 3-week treatment interval] or infusion #3 [for 4-week treatment interval]; SC: before last SC infusion) 60 minutes pre-infusion up to 28 days (+/-2 days) post-infusion
Population: Participants ≥ 12 years exposed to either or both study drugs with PK measurements at the following time points: Pre-infusion and 30-minutes post-infusion (Day 0) IV- Days 1, 4, 9, 14, 21, 28* SC- Days 1, 3, 5, 9, 14, 21, 28* *Measurements at Day 28 for the 4-week treatment interval only
Measure: Median (95% Confidence Interval); unit: g/L
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 68 | 60
g/L | 10.1 [9.5 to 10.9] | 10.4 [9.4 to 11.2]

13. Secondary Outcome: IgG Area Under the Curve (AUC)/Week for Participants Aged 12 Years and Older
Description: Immunoglobulin (IgG) Area under the Curve (AUC) AUC/week after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older. The AUC between adjacent infusions was calculated by the trapezoidal rule. Linear interpolation/extrapolation was used to calculate the AUC for the exact duration of the infusion intervals (21 days for 3-week treatment interval or 28 days for 4-week treatment interval).
Time Frame: PK evaluations: (IV: before infusion #4 [for 3-week treatment interval] or infusion #3 [for 4-week treatment interval];SC: before last SC infusion) 60 minutes pre-infusion up to 28 days (+/-2 days) post-infusion.
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: g*days/L
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 68 | 60
g*days/L | 93.9 [89.1 to 102.1] | 90.5 [83.8 to 98.4]

14. Secondary Outcome: IgG Clearance (CL) for Participants Aged 12 Years and Older
Description: Immunoglobulin (IgG) Clearance after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older. Clearance (CL) is provided after administration of IGIV,10% given via IV route. Apparent Clearance is provided after administration of IGIV, 10% given via SC route with rHuPH20. Clearance and apparent clearance are determined by weight adjusted dose divided by total AUC.
Time Frame: as for outcome 13
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: mL/kg/day
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 68 | 60
mL/kg/day | 1.4 [1.2 to 1.4] | 1.6 [1.4 to 1.7]

15. Secondary Outcome: IgG Maximum Plasma Concentration (C_max) for Participants Aged 12 Years and Older
Description: Maximum immunoglobulin (IgG) concentration after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: g/L
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 68 | 60
g/L | 21.9 [20.7 to 23.9] | 15.5 [14.5 to 17.1]

16. Secondary Outcome: IgG Terminal Half Life (T1/2) for Participants Aged 12 Years and Older
Description: Terminal half life (T1/2) for immunoglobulin (IgG) after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older. Terminal half life is the time it takes for the plasma concentration or the amount of immunoglobulin in the body to be reduced by 50% during the terminal phase
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 68 | 60
Days | 35.7 [32.4 to 40.4] | 45.3 [41.0 to 60.2]

17. Secondary Outcome: Time to Maximum IgG Concentration (T-max) for Participants Aged 12 Years and Older
Description: Time to Maximum Immunoglobulin (IgG) Concentration (T-max) after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 68 | 60
Days | 0.1 [0.1 to 0.1] | 5.0 [3.3 to 5.1]

18. Secondary Outcome: Tetanus Antibody Minimum Plasma Concentration (C_min) for Participants Aged 12 Years and Older
Description: Minimal tetanus (clostridium tetani toxoid) antibody concentration after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: IU/mL
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 46 | 60
IU/mL | 2.3 [2.2 to 2.7] | 2.1 [1.9 to 2.4]

19. Secondary Outcome: Tetanus Antibody Area Under the Curve (AUC)/Week for Participants Aged 12 Years and Older
Description: Tetanus (clostridium tetani toxoid) antibody Area under the Curve (AUC) AUC/week after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older. The AUC between adjacent infusions was calculated by the trapezoidal rule. Linear interpolation/extrapolation was used to calculate the AUC for the exact duration of the infusion intervals (21 days for 3-week treatment interval or 28 days for 4-week treatment interval).
Time Frame: as for outcome 13
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: IU*days/mL
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 46 | 60
IU*days/mL | 28.0 [27.0 to 32.2] | 22.6 [19.9 to 25.6]

20. Secondary Outcome: Tetanus Antibody Clearance (CL) for Participants Aged 12 Years and Older
Description: Tetanus (clostridium tetani toxoid) antibody Clearance after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older. Clearance (CL) is provided after administration of IGIV,10% given via IV route. Apparent Clearance is provided after administration of IGIV, 10% given via SC route with rHuPH20. Clearance (CL) and apparent clearance are determined by weight adjusted dose divided by total AUC.
Time Frame: as for outcome 13
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: nL/IU/day
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 46 | 60
nL/IU/day | 4.5 [3.9 to 5.1] | 5.8 [5.4 to 7.0]

21. Secondary Outcome: Tetanus Antibody Terminal Half Life (T1/2) for Participants Aged 12 Years and Older
Description: Terminal half life (T1/2) for tetanus (clostridium tetani toxoid) antibody after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older. Terminal half life is the time it takes for the plasma concentration or the amount of tetanus antibody in the body to be reduced by 50% during the terminal phase
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 44 | 50
Days | 22.7 [20.0 to 28.1] | 30.4 [25.7 to 37.2]

22. Secondary Outcome: Tetanus Antibody Maximum Plasma Concentration (C_max) for Participants Aged 12 Years and Older
Description: Maximum tetanus (clostridium tetani toxoid) antibody concentration after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: IU/mL
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 46 | 60
IU/mL | 7.3 [6.8 to 8.1] | 5.0 [4.4 to 5.6]

23. Secondary Outcome: Time to Maximum Tetanus Antibody Concentration (T-max) for Participants Aged 12 Years and Older
Description: Time to Maximum tetanus (clostridium tetani toxoid) antibody Concentration (T-max) after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 46 | 60
Days | 0.1 [0.1 to 0.2] | 5.1 [4.0 to 6.0]

24. Secondary Outcome: H. Influenzae Antibody Minimum Plasma Concentration (C_min) for Participants Aged 12 Years and Older
Description: Minimal influenza (haemophilus influenzae) antibody concentration after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: μg/mL
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 46 | 60
μg/mL | 2.1 [2.0 to 2.6] | 2.2 [1.8 to 2.6]

25. Secondary Outcome: H. Influenzae Antibody Area Under the Curve (AUC)/Week for Participants Aged 12 Years and Older
Description: Influenza (haemophilus influenzae) antibody Area under the Curve (AUC) AUC/week after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older. The AUC between adjacent infusions was calculated by the trapezoidal rule. Linear interpolation/extrapolation was used to calculate the AUC for the exact duration of the infusion intervals (21 days for 3-week treatment interval or 28 days for 4-week treatment interval).
Time Frame: as for outcome 13
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: μg*days/mL
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 46 | 60
μg*days/mL | 22.4 [21.1 to 26.6] | 22.5 [20.8 to 24.3]

26. Secondary Outcome: H. Influenzae Antibody Clearance (CL) for Participants Aged 12 Years and Older
Description: Influenza (haemophilus influenzae) antibody Clearance after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older. Clearance (CL) is provided after administration of IGIV,10% given via IV route. Apparent Clearance is provided after administration of IGIV, 10% given via SC route with rHuPH20. Clearance (CL) and apparent clearance are determined by weight adjusted dose divided by total AUC.
Time Frame: as for outcome 13
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: L/kg/day
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 46 | 60
L/kg/day | 5.8 [5.3 to 6.5] | 6.4 [5.8 to 7.1]

27. Secondary Outcome: H. Influenzae Antibody Maximum Plasma Concentration (C_max) for Participants Aged 12 Years and Older
Description: Maximal influenza (haemophilus influenzae) antibody concentration after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: μg/mL
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 46 | 60
μg/mL | 5.5 [5.1 to 6.8] | 4.1 [3.8 to 4.5]

28. Secondary Outcome: H. Influenzae Antibody Terminal Half Life (T1/2) for Participants Aged 12 Years and Older
Description: Terminal half life (T1/2) for influenza (haemophilus influenzae) antibody after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older. Terminal half life is the time it takes for the plasma concentration or the amount of influenza antibody in the body to be reduced by 50% during the terminal phase.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 45 | 55
Days | 33.8 [25.6 to 45.3] | 35.0 [32.3 to 41.0]

29. Secondary Outcome: Time to Maximum H. Influenzae Antibody Concentration (T-max) for Participants Aged 12 Years and Older
Description: Time to Maximum influenza (haemophilus influenzae) antibody Concentration (T-max) after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) for participants aged 12 years and older
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 46 | 60
Days | 0.1 [0.1 to 0.2] | 4.8 [3.3 to 5.0]

30. Secondary Outcome: Rate of Days Off School or Work
Description: Monthly rate of days off school or work after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up. Point estimates and 95% CIs for the monthly rates were calculated using a Poisson model and the same methodology including allowance for over-dispersion as described for the primary outcome measures. The lengths of the month were defined as average length of the month in the Gregorian calendar, namely (365*400+100-3)/(400*12)= 30.436875 days.
Time Frame: Monthly, for up to 17 months
Population: Full Analysis Data Set
Measure: Number (95% Confidence Interval); unit: Days off per month
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 81 | 81
Days off per month | 0.23 [0.15 to 0.34] | 0.28 [0.20 to 0.37]

31. Secondary Outcome: Rate of Days on Antibiotics
Description: Monthly rate of days on antibiotics after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up. Point estimates and 95% CIs for the monthly rates were calculated using a Poisson model and the same methodology including allowance for over-dispersion as described for the primary outcome measures. The lengths of the month was defined as average length of the month in the Gregorian calendar, namely (365*400+100-3)/(400*12)= 30.436875 days.
Time Frame: Monthly, for up to 17 months
Population: Full Analysis Data Set
Measure: Number (95% Confidence Interval); unit: Days on antibiotics per month
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 81 | 81
Days on antibiotics per month | 3.15 [2.19 to 4.35] | 1.69 [1.29 to 2.16]

32. Secondary Outcome: Rate of Acute Physician Visits
Description: Monthly rate of acute physician visits after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up. Point estimates and 95% CIs for the monthly rates will be calculated using a Poisson model and the same methodology including allowance for over-dispersion as described for the primary outcome measures. The lengths of the month will be defined as average length of the month in the Gregorian calendar, namely (365*400+100-3)/(400*12)= 30.436875 days.
Time Frame: Monthly, for up to 17 months
Population: Full Analysis Data Set
Measure: Number (95% Confidence Interval); unit: Visits per month
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 81 | 81
Visits per month | 0.33 [0.23 to 0.45] | 0.40 [0.32 to 0.49]

33. Secondary Outcome: Rate of Days in Hospital
Description: Monthly rate of days in hospital after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up. Point estimates and 95% CIs for the monthly rates will be calculated using a Poisson model and the same methodology including allowance for over-dispersion as described for the primary outcome measures. The lengths of the month will be defined as average length of the month in the Gregorian calendar, namely (365*400+100-3)/(400*12)= 30.436875 days.
Time Frame: Monthly, for up to 17 months
Population: Full Analysis Data Set
Measure: Number (95% Confidence Interval); unit: Days per month
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 81 | 81
Days per month | 0.06 [0.03 to 0.10] | 0.02 [0.01 to 0.03]

34. Secondary Outcome: Percentage of Participants for Which the Infusion Rate Was Reduced and/or the Infusion Interrupted or Stopped for Tolerability Concerns or for Adverse Events (AEs)
Description: Percentage of participants for which the infusion rate was reduced and/or the infusion interrupted or stopped during administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up for tolerability concerns or for adverse events (AEs). An infusion was deemed as tolerated if there are no serious Adverse Drug Reactions (ADR), no non-serious moderate or severe local ADRs that prevent completion of the infusion and no non-serious moderate or severe systemic ADRs during infusion or within 60 minutes of completion of the infusion.
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Percentage of participants
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Percentage of participants
  % participants with reduced infusion rate only | 6.9 | 9.9
  % participants with interrupted infusion rate only | 4.6 | 4.9
  % participants with infusion stopped only | 0.0 | 1.2
  % participants with no changes to infusion rate | 88.5 | 84.0

35. Secondary Outcome: Percentage of Infusions for Which the Infusion Rate Was Reduced and/or the Infusion Interrupted or Stopped for Tolerability Concerns or for Adverse Events (AEs)
Description: Percentage of infusions for which the infusion rate was reduced and/or the infusion interrupted or stopped during administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up for tolerability concerns or for adverse events (AEs). IV administration of IGIV, 10%: 365 infusions; SC administration of IGIV, 10% with rHuPH20: 1129 infusions
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Percentage of infusions
  % infusions with infusion rate reduced only | 2.7 | 1.7
  % infusions with interrupted infusion rate only | 1.4 | 0.4
  % infusions with infusion stopped only | 0.0 | 0.2
  % infusions with no changes to infusion rate | 95.9 | 97.7

36. Secondary Outcome: Rate of Temporally Associated AEs Per Infusion
Description: Rate of all AEs (including and excluding infections) per infusion that began during administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up (during infusion) or within 72 hours of completion of an infusion ("temporally associated")
Time Frame: During infusion or within 72 hours of completion of infusion
Population: Safety Analysis Data Set (SADS)
Measure: Median (95% Confidence Interval); unit: Number of AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Number of AEs per infusion
  Including infections | 0.25 [0.20 to 0.50] | 0.21 [0.13 to 0.31]
  Excluding infections | 0.25 [0.20 to 0.40] | 0.17 [0.09 to 0.26]

37. Secondary Outcome: Percentage of Participants Reporting ≥1 Temporally Associated AEs
Description: Percentage of participants reporting at least 1 AE (including and excluding infections) during administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up (during infusion) or within 72 hours of completion of infusion ("temporally associated")
Time Frame: During infusion or within 72 hours of completion of infusion
Population: Safety Analysis Data Set
Measure: Number; unit: Percentage of participants
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Percentage of participants
  Including infections | 66.7 | 86.4
  Excluding infections | 63.2 | 82.7

38. Secondary Outcome: Percentage of Infusions Resulting in ≥1 Temporally Associated AEs
Description: Percentage of infusions resulting in at least 1 AE (including and excluding infections) during administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up (during infusion) or within 72 hours of completion of infusion ("temporally associated")
Time Frame: During infusion or within 72 hours of completion of infusion
Population: Safety Analysis Data Set
Measure: Number; unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Percentage of infusions
  Including infections | 30.1 | 24.5
  Excluding infections | 28.8 | 22.8

39. Secondary Outcome: Percentage of Participants Reporting ≥1 Temporally Associated Moderate or Severe AEs
Description: Percentage of participants reporting at least 1 Moderate or Severe AE (including and excluding infections) during administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up (during infusion) or within 72 hours of completion of infusion ("temporally associated")
Time Frame: During infusion or within 72 hours of completion of infusion
Population: Safety Analysis Data Set
Measure: Number; unit: Percentage of participants
Groups:
- SC Administration of IGIV, 10% With rHuPH20 Including Ramp-up: Includes 2 participants who withdrew during ramp-up SC and rHuPH20 administration of IGIV, 10%
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 Including Ramp-up
Number analyzed (Participants) | 87 | 83
Percentage of participants
  Including infections | 36.8 | 54.3
  Excluding infections | 34.5 | 46.9

40. Secondary Outcome: Percentage of Infusions Resulting in ≥1 Temporally Associated Moderate or Severe AEs Within 72 Hours of Completion of Infusion
Description: Percentage of infusions resulting in at least 1 moderate or severe AE (including and excluding infections) during administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up (during infusion) or within 72 hours of completion of infusion ("temporally associated")
Time Frame: During infusion or within 72 hours of completion of infusion
Population: Safety Analysis Data Set
Measure: Median (95% Confidence Interval); unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Percentage of infusions
  Including infections | 0.0 [0.0 to 0.0] | 5.9 [0.0 to 7.1]
  Excluding infections | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 6.3]

41. Secondary Outcome: Percentage of SC Doses of IGIV, 10% and rHuPH20 Tolerated at 1 Infusion Site
Description: Percentage of subcutaneous (SC) doses of immune globulin intravenous (IGIV), 10% and recombinant human hyaluronidase (rHuPH20) tolerated at 1 infusion site. An infusion was deemed as tolerated if there were no serious adverse drug reactions (ADRs), no non-serious moderate or severe local ADRs that prevented completion of the infusion, and no non-serious moderate or severe systemic ADRs during or within 60 minutes of completion of the infusion.
Time Frame: During infusion or within 60 minutes of completion of the infusion
Population: Safety Analysis Data Set
Measure: Median (95% Confidence Interval); unit: Percentage of infusions
Groups:
- SC Administration of IGIV, 10% With rHuPH20 at Ramp-up: At start of SC administration of IGIV, 10% with rHuPH20, the first SC dose was a 1-week dose given for a 1-week interval, then if the 1 week SC infusions were tolerated, each week the interval (and dose) was increased by 1 week, until the treatment interval was the same as the interval for intravenous treatment (3 weeks or 4 weeks)
Arm/Group | SC Administration of IGIV, 10% With rHuPH20 at Ramp-up | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 83 | 81
Percentage of infusions | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

42. Secondary Outcome: Percentage of Infusions Associated With ≥1 Systemic AE During Infusion or Within 72 Hours of Completion of Infusion
Description: Percentage of intravenous (IV) and subcutaneous (SC) infusions associated with ≥1 systemic AE (including and excluding infections) during administration of immune globulin intravenous (IGIV), 10% given via IV or SC route with recombinant human hyaluronidase (rHuPH20) after ramp-up (during infusion) or within 72 hours of completion of infusion
Time Frame: During infusion or within 72 hours of completion of infusion
Population: Safety Analysis Data Set
Measure: Median (95% Confidence Interval); unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Percentage of infusions
  Including infections | 25.0 [20.0 to 25.0] | 8.3 [7.7 to 12.5]
  Excluding infections | 25.0 [16.7 to 25.0] | 8.3 [6.3 to 10.0]

43. Secondary Outcome: Percentage of Participants With ≥1 Systemic AE (Including and Excluding Infections) During Infusion or Within 72 Hours of Completion of Infusion
Description: Percentage of participants with ≥1 systemic AE (including and excluding Infections) during administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up (during infusion) or within 72 hours of completion of infusion
Time Frame: During infusion or within 72 hours of completion of infusion
Population: Participants exposed to either or both study drugs
Measure: Number; unit: Percentage of participants
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Percentage of participants
  Including infections | 64.4 | 75.3
  Excluding infections | 60.9 | 67.9

44. Secondary Outcome: Percentage of Infusions Associated With ≥1 Local AE (Including and Excluding Infections) During Infusion or Within 72 Hours of Completion of Infusion
Description: Percentage of IV and SC (with recombinant human hyaluronidase [rHuPH20]) infusions associated with ≥1 local AE (including and excluding infections) during administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with rHuPH20 after ramp-up (during infusion) or within 72 hours of completion of infusion
Time Frame: During infusion or within 72 hours of completion of infusion
Population: Safety Analysis Data Set
Measure: Median (95% Confidence Interval); unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Percentage of infusions
  Including infections | 0.0 [0.0 to 0.0] | 5.9 [0.0 to 8.3]
  Excluding infections | 0.0 [0.0 to 0.0] | 5.9 [0.0 to 8.3]

45. Secondary Outcome: Percentage of Infusions Associated With ≥1 Local AE At Any Time During the Study
Description: Percentage of intravenous (IV) and subcutaneous (SC) infusions with recombinant human hyaluronidase (rHuPH20) after ramp-up of immune globulin intravenous (IGIV), 10% associated with ≥1 local AE (including and excluding infections) at any time during the study
Time Frame: At any time during the study
Population: Safety Analysis Data Set
Measure: Median (95% Confidence Interval); unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Percentage of infusions
  Including infections | 0.0 [0.0 to 0.0] | 5.9 [0.0 to 8.3]
  Excluding infections | 0.0 [0.0 to 0.0] | 5.9 [0.0 to 8.3]

46. Secondary Outcome: Percentage of Participants With ≥1 Local AE During Infusion or Within 72 Hours of Completion of Infusion
Description: Percentage of participants With ≥1 local AE (including and excluding Infections) during administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up (during infusion) or within 72 hours of completion of infusion
Time Frame: During infusion or within 72 hours of completion of infusion
Population: Safety Analysis Data Set
Measure: Number; unit: Percentage of participants
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Percentage of participants
  Including infections | 4.6 | 51.9
  Excluding infections | 4.6 | 51.9

47. Secondary Outcome: Percentage of Participants With ≥1 Local AE At Any Time During the Study
Description: Percentage of participants With ≥1 local AE (including and excluding infections) after administration of immune globulin intravenous (IGIV), 10% given via intravenous (IV) or subcutaneous (SC) route with recombinant human hyaluronidase (rHuPH20) after ramp-up at any time during the study
Time Frame: During infusion or within 72 hours of completion of infusion
Population: Safety Analysis Data Set
Measure: Number; unit: Percentage of participants
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Percentage of participants
  Including infections | 5.7 | 53.1
  Excluding infections | 5.7 | 53.1

48. Secondary Outcome: Rate of AEs Determined to be Related to the Study Drug by the Investigator Per Participant
Description: Rate of related AEs defined as the total number of AEs determined by the investigator to be related to the study drug (immune globulin intravenous [IGIV], 10% or recombinant human hyaluronidase [rHuPH20]), that occur at any time during the study divided by the total number of participants
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Median (95% Confidence Interval); unit: Number of AEs per participant
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 Including Ramp-up
Number analyzed (Participants) | 87 | 81
Number of AEs per participant
  Including infections | 0.00 [0.00 to 0.25] | 0.09 [0.07 to 0.25]
  Excluding infections | 0.00 [0.00 to 0.25] | 0.09 [0.07 to 0.25]

49. Secondary Outcome: Rate of AEs Determined to be Related to the Study Drug by the Investigator Per Infusion
Description: Rate of related AEs defined as the total number of AEs determined by the investigator to be related to the study drug (immune globulin intravenous [IGIV], 10% or recombinant human hyaluronidase [rHuPH20]), that occur at any time during the study divided by the total number of infusions
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Median (95% Confidence Interval); unit: Number of AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Number of AEs per infusion
  Including infections | 0.25 [0.25 to 0.50] | 0.22 [0.13 to 0.31]
  Excluding infections | 0.25 [0.20 to 0.50] | 0.18 [0.12 to 0.26]

50. Secondary Outcome: Frequency of Dose Corrections (If IgG Trough Levels <4.5 g/L) for Each Study Epoch (IV and SC/rHuPH20 Treatment)
Description: Frequency of dose corrections based on immune globulin G (IgG) trough levels <4.5 g/L IgG, if any, for intravenous (IV) (Epoch 1) and subcutaneous with recombinant human hyaluronidase (SC/rHuPH20) after ramp-up (Epoch 2) administration of immune globulin intravenous (IGIV), 10% Defined/calculated as the number of participants requiring dose adjustments divided by the number of participants, for each respective data set.
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Percentage of participants
Groups:
- Study Epoch 1: Epoch 1 - IV administration of IGIV, 10%
- Study Epoch 2: Epoch 2 - SC administration of IGIV, 10% with rHuPH20 after ramp-up
Arm/Group | Study Epoch 1 | Study Epoch 2
Number analyzed (Participants) | 87 | 81
Percentage of participants | 0.0 | 0.0

51. Secondary Outcome: Number of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to Study Drug, and Severity (A-F)
Description: Categories presented as Preferred term-Seriousness, Relatedness, Severity. The following codes are to be used: Seriousness: non-SAE-non-serious AE; SAE-serious AE Relationship: NR-not related to immune globulin (IGIV), 10% and recombinant human hyaluronidase (rHuPH20); RIGIV-related to IGIV, 10%; RrHu-related to rHuPH20; Rboth-related to both IGIV, 10% and rHuPH20 Severity: Mild; Mod (Moderate); Severe Preferred terms abbreviated: ADHD-Attention Deficit/Hyperactivity Disorder BP-Blood Pressure COPD- Chronic Obstructive Pulmonary Disease
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number of AEs
  Abdominal Discomfort-non-SAE, NR, Mod | 0 | 1
  Abdominal Distension-non-SAE, Rboth, Mild | 0 | 1
  Abdominal Hernia-non-SAE, NR, Mild | 0 | 1
  Abdominal Pain-non-SAE, NR, Mild | 1 | 2
  Abdominal Pain-non-SAE, NR, Mod | 0 | 1
  Abdominal Pain-non-SAE, Rboth, Mild | 0 | 3
  Abdominal Pain-non-SAE, Rboth, Mod | 0 | 1
  Abdominal Pain Lower-non-SAE, NR, Mild | 0 | 1
  Abdominal Pain Upper-non-SAE, NR, Mild | 1 | 5
  Abdominal Pain Upper-non-SAE, NR, Mod | 1 | 0
  Abdominal Pain Upper-non-SAE, RIGIV, Mild | 0 | 1
  Abdominal Pain Upper-non-SAE, RIGIV, Mod | 1 | 0
  Abdominal Pain Upper-non-SAE, Rboth, Mild | 0 | 2
  Abdominal Tenderness-non-SAE, NR, Mod | 1 | 0
  Abdominal Tenderness-non-SAE, RIGIV, Mild | 0 | 1
  Abdominal Tenderness-non-SAE, RIGIV, Mod | 0 | 2
  Acarodermatitis-non-SAE, NR, Mild | 0 | 1
  Acne-non-SAE, NR, Mild | 1 | 1
  Acute Sinusitis-non-SAE, NR, Mild | 1 | 0
  Acute Sinusitis-non-SAE, NR, Mod | 0 | 4
  Adenoidal Hypertrophy-non-SAE, NR, Mod | 0 | 1
  Adnexa Uteri Cyst-non-SAE, NR, Mild | 1 | 0
  Adrenocortical Insufficiency Acute-SAE, NR, Mod | 0 | 1
  Allergic Respiratory Symptom-non-SAE, NR, Mild | 0 | 1
  Allergic Sinusitis-non-SAE, NR, Mild | 1 | 0
  Alopecia-non-SAE, NR, Mild | 1 | 0
  Animal Bite-non-SAE, NR, Mod | 1 | 0
  Antibody Test Positive-non-SAE, Rboth, Mod | 0 | 1
  Anxiety-non-SAE, NR, Mild | 0 | 1
  Anxiety-non-SAE, NR, Mod | 1 | 0
  Aphthous Stomatitis-non-SAE, NR, Mild | 2 | 1
  Aphthous Stomatitis-non-SAE, NR, Mod | 0 | 1
  Arteriosclerosis Coronary Artery-non-SAE, NR, Mild | 0 | 1
  Arthralgia-non-SAE, NR, Mild | 0 | 5
  Arthralgia-non-SAE, NR, Mod | 1 | 6
  Arthralgia-non-SAE, RIGIV, Mild | 0 | 1
  Arthralgia-non-SAE, RIGIV, Mod | 0 | 2
  Arthritis-non-SAE, NR, Mod | 1 | 1
  Arthropathy-non-SAE, NR, Mod | 1 | 0
  Arthropod Bite-non-SAE, NR, Mild | 2 | 2
  Arthropod Sting-non-SAE, NR, Mild | 0 | 1
  Arthropod Sting-non-SAE, NR, Mod | 1 | 0
  Aspiration-non-SAE, NR, Mild | 0 | 1
  Asthenia-non-SAE, NR, Mild | 0 | 3
  Asthenia-non-SAE, NR, Mod | 1 | 0
  Asthenia-non-SAE, RIGIV, Mild | 0 | 1
  Asthma-non-SAE, NR, Mild | 0 | 4
  Asthma-non-SAE, NR, Mod | 8 | 21
  Asthma-non-SAE, NR, Severe | 0 | 1
  ADHD-non-SAE, NR, Mod | 0 | 1
  Back Injury-non-SAE, NR, Mod | 1 | 0
  Back Injury-SAE, NR, Severe | 0 | 1
  Back Pain-non-SAE, NR, Mild | 1 | 2
  Back Pain-non-SAE, NR, Mod | 1 | 5
  Bacterial Prostatitis-non-SAE, NR, Mild | 0 | 1
  Blepharitis-non-SAE, NR, Mod | 1 | 0
  Blister-non-SAE, NR, Mild | 0 | 1
  Blood Pressure Decreased-non-SAE, NR, Mild | 0 | 1
  Blood Pressure Decreased-non-SAE, Rboth, Mild | 0 | 1
  Blood Pressure Increased-non-SAE, NR, Mod | 0 | 1
  Blood Pressure Increased-non-SAE, RIGIV, Mild | 0 | 1
  Blood Pressure Increased-non-SAE, RIGIV, Mod | 0 | 1
  Blood Pressure Increased-non-SAE, RrHu, Mild | 0 | 1
  BP Systolic Increased-non-SAE, RIGIV, Mild | 1 | 0
  Blood Urea Increased-non-SAE, NR, Mild | 0 | 1
  Body Fat Disorder-non-SAE, NR, Mild | 0 | 1
  Body Tinea-non-SAE, NR, Mild | 1 | 0
  Body Tinea-non-SAE, NR, Mod | 0 | 1
  Bone Pain-non-SAE, NR, Mild | 0 | 1
  Breast Pain-non-SAE, NR, Mild | 1 | 0
  Bronchal Hyperreactivity-non-SAE, NR, Mild | 0 | 1
  Bronchitis-non-SAE, NR, Mild | 4 | 2
  Bronchitis-non-SAE, NR, Mod | 2 | 8
  Bronchitis-SAE, NR, Mod | 1 | 0
  Bronchospasm-non-SAE, NR, Mod | 0 | 1
  Burn Infection-non-SAE, NR, Mild | 0 | 1
  Burning Sensation-non-SAE, RIGIV, Mild | 0 | 1
  Burning Sensation-non-SAE, RIGIV, Mod | 0 | 1
  Burning Sensation-non-SAE, RrHu, Mild | 0 | 1
  Bursitis-non-SAE, NR, Mild | 1 | 0
  Bursitis-non-SAE, NR, Mod | 0 | 1
  Candidiasis-non-SAE, NR, Mild | 1 | 0
  Candidiasis-non-SAE, NR, Mod | 1 | 1
  Cardiac Murmur-non-SAE, NR, Mild | 0 | 1
  Cellulitis-non-SAE, NR, Mild | 0 | 1
  Cellulitis-non-SAE, NR, Mod | 0 | 3
  Cellulitis-non-SAE, Rboth, Mod | 0 | 1
  Cerumen Impaction-non-SAE, NR, Mild | 0 | 2
  Cervical Dysplasia-SAE, NR, Mild | 1 | 1
  Cheilitis-non-SAE, NR, Mild | 2 | 0
  Chest Pain-non-SAE, NR, Mild | 0 | 2
  Chills-non-SAE, NR, Mild | 0 | 3
  Chills-non-SAE, RIGIV, Mild | 6 | 1
  Chills-non-SAE, RIGIV, Mod | 3 | 0
  Chills-non-SAE, Rboth, Mild | 0 | 1
  COPD-non-SAE, NR, Mod | 0 | 2
  COPD-non-SAE, NR, Severe | 1 | 0
  Chronic Sinusitis-non-SAE, NR, Mild | 0 | 4
  Chronic Sinusitis-non-SAE, NR, Mod | 1 | 1
  Concussion-non-SAE, NR, Mod | 1 | 0
  Confusional State-non-SAE, NR, Mod | 0 | 1
  Confusional State-non-SAE, RIGIV, Mild | 1 | 0
  Conjunctivitis-non-SAE, NR, Mild | 1 | 2
  Conjunctivitis Allergic-non-SAE, NR, Mild | 1 | 0
  Conjunctivitis Allergic-non-SAE, NR, Mod | 1 | 0
  Conjunctivitis Bacterial-non-SAE, NR, Mild | 1 | 1
  Conjunctivitis Bacterial-non-SAE, NR, Mod | 0 | 1
  Conjunctivitis Bacterial-non-SAE, NR, Severe | 0 | 1
  Constipation-non-SAE, NR, Mild | 0 | 3
  Contusion-non-SAE, NR, Mild | 1 | 5
  Contusion-non-SAE, NR, Mod | 1 | 0
  Contusion-non-SAE, RIGIV, Mod | 0 | 1
  Coombs Test Positive-non-SAE, RIGIV, Mild | 0 | 1
  Costochondritis-non-SAE, NR, Mod | 0 | 1
  Cough-non-SAE, NR, Mild | 3 | 6
  Cough-non-SAE, NR, Mod | 0 | 2
  Cough-non-SAE, RIGIV, Mild | 1 | 0
  Cushingoid-non-SAE, NR, Mild | 0 | 1
  Cystitis-non-SAE, NR, Mild | 0 | 1
  Deafness Neurosensory-non-SAE, NR, Mild | 1 | 0
  Decreased Appetite-non-SAE, NR, Mild | 1 | 1
  Decreased Appetite-non-SAE, RrHu, Mild | 0 | 1
  Decreased Appetite-non-SAE, Rboth, Mild | 0 | 2
  Dehydration-non-SAE, NR, Mod | 0 | 2
  Dental Caries-non-SAE, NR, Mild | 0 | 2
  Dental Caries-non-SAE, NR, Mod | 0 | 3
  Depressed Mood-non-SAE, NR, Mild | 0 | 1
  Depression-non-SAE, NR, Severe | 0 | 1
  Dermal Cyst-non-SAE, NR, Mild | 0 | 1
  Dermatitis-non-SAE, NR, Mild | 0 | 2
  Dermatitis-non-SAE, NR, Mod | 1 | 0
  Dermatitis Acneiform-non-SAE, NR, Mod | 1 | 0
  Dermatitis Contact-non-SAE, NR, Mild | 0 | 2
  Dermatitis Contact-non-SAE, NR, Mod | 2 | 2
  Dermatitis Infected-non-SAE, NR, Mild | 0 | 2
  Dermatitis Infected-non-SAE, NR, Mod | 0 | 1
  Dermatitis Infected-non-SAE, NR, Severe | 0 | 1
  Device Failure-non-SAE, NR, Mild | 2 | 1
  Device Failure-non-SAE, NR, Mod | 0 | 2
  Diarrhoea-non-SAE, NR, Mild | 3 | 6
  Diarrhoea-non-SAE, NR, Mod | 2 | 4
  Diarrhoea-non-SAE, RIGIV, Mild | 1 | 1
  Diarrhoea-non-SAE, RIGIV, Mod | 1 | 0
  Diarrhoea Haemorrhagic-non-SAE, NR, Mild | 1 | 0
  Diarrhoea Infectious-non-SAE, NR, Mild | 0 | 1
  Diastolic Dysfunction-non-SAE, NR, Mild | 0 | 1
  Disaccharide Metabolism Disorder-non-SAE, NR, Mild | 0 | 1
  Disturbance in Attention-non-SAE, NR, Mild | 0 | 2
  Diverticulitis-non-SAE, NR, Mod | 1 | 0
  Dizziness-non-SAE, NR, Mild | 2 | 7
  Dizziness-non-SAE, NR, Mod | 0 | 2
  Dizziness-non-SAE, RIGIV, Mild | 0 | 3
  Dizziness-non-SAE, RIGIV, Mod | 1 | 0
  Drug Eruption-non-SAE, NR, Mod | 1 | 0
  Dry Eye-non-SAE, NR, Mod | 0 | 1
  Dry Mouth-non-SAE, NR, Mild | 0 | 1
  Dry Skin-non-SAE, NR, Mild | 0 | 3
  Dysmenorrhoea-non-SAE, NR, Mild | 0 | 1
  Dyspepsia-non-SAE, NR, Mild | 0 | 2
  Dyspepsia-non-SAE, NR, Mod | 0 | 1
  Dyspepsia-non-SAE, RIGIV, Mild | 1 | 0
  Dysphagia-non-SAE, NR, Mild | 0 | 1
  Dysphagia-non-SAE, NR, Mod | 0 | 1
  Dyspnoea-non-SAE, NR, Mild | 1 | 0
  Dyspnoea-non-SAE, NR, Mod | 1 | 0
  Dyspnoea-non-SAE, RIGIV, Mild | 1 | 0
  Dysuria-non-SAE, NR, Mild | 0 | 2
  Ear Infection-non-SAE, NR, Mild | 2 | 2
  Ear Infection-non-SAE, NR, Mod | 1 | 1
  Ear Pain-non-SAE, NR, Mild | 3 | 2
  Ear Pain-non-SAE, NR, Mod | 0 | 1
  Ecchymosis-non-SAE, NR, Mild | 0 | 1
  Eczema-non-SAE, NR, Mild | 0 | 1
  Eczema-non-SAE, NR, Mod | 0 | 1
  Eczema-non-SAE, NR, Severe | 1 | 0
  Eosinophil Count-non-SAE, NR, Mild | 0 | 1
  Epitaxis-non-SAE, NR, Mild | 2 | 3
  Epitaxis-non-SAE, NR, Mod | 2 | 2
  Erythema-non-SAE, NR, Mild | 1 | 0
  Erythema-non-SAE, RIGIV, Mod | 0 | 1
  Erythema-non-SAE, RrHu, Mild | 0 | 1
  Erythema-non-SAE, Rboth, Mild | 0 | 1
  Erythema-non-SAE, Rboth, Mod | 0 | 1
  Eustachian Tube Dysfunction-non-SAE, NR, Mild | 1 | 0
  Excoriation-non-SAE, NR, Mild | 2 | 2
  Extravasation Blood-non-SAE, Rboth, Mild | 0 | 1
  Eye Irritation-non-SAE, NR, Mild | 0 | 1
  Eye Pruritus-non-SAE, NR, Mod | 0 | 1
  Eye Swelling-non-SAE, NR, Mod | 0 | 1
  Fall-non-SAE, NR, Mild | 0 | 1
  Fall-non-SAE, NR, Mod | 0 | 1
  Fatigue-non-SAE, NR, Mild | 1 | 5
  Fatigue-non-SAE, NR, Mod | 1 | 2
  Fatigue-non-SAE, RIGIV, Mild | 8 | 8
  Fatigue-non-SAE, RIGIV, Mod | 0 | 3
  Fatigue-non-SAE, Rboth, Mild | 0 | 3
  Feeling Abnormal-non-SAE, Rboth, Mod | 0 | 1
  Feeling Cold-non-SAE, RIGIV, Mild | 2 | 0
  Flatulence-non-SAE, NR, Mild | 0 | 1
  Flatulence-non-SAE, NR, Mod | 0 | 1
  Food Poisoning-non-SAE, NR, Mod | 0 | 1
  Free Haemoglobin Present-non-SAE, NR, Mild | 1 | 1
  Free Haemoglobin Present-non-SAE, NR, Severe | 1 | 0

52. Secondary Outcome: Number of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to Study Drug, and Severity (G-M)
Description: Categories presented as Preferred term-Seriousness, Relatedness, Severity. The following codes are to be used: Seriousness: non-SAE-non-serious AE; SAE-serious AE Relationship: NR-not related to immune globulin (IGIV), 10% and recombinant human hyaluronidase (rHuPH20); RIGIV-related to IGIV, 10%; RrHu-related to rHuPH20; Rboth-related to both IGIV, 10% and rHuPH20 Severity: Mild; Mod (Moderate); Severe
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number of AEs
  Gait Disturbance-non-SAE, NR, Mild | 0 | 1
  Gastroenteritis-non-SAE, NR, Mild | 0 | 3
  Gastroenteritis-non-SAE, NR, Mod | 2 | 2
  Gastroenteritis-non-SAE, RIGIV, Mild | 1 | 0
  Gastroenteritis-SAE, NR, Mod | 0 | 1
  Gastroenteritis Bacterial-non-SAE, NR, Mod | 0 | 1
  Gastroenteritis Viral-non-SAE, NR, Mild | 3 | 6
  Gastroenteritis Viral-non-SAE, NR, Mod | 0 | 5
  Gastroenteritis Viral-non-SAE, RIGIV, Mild | 0 | 1
  Gastrointestinal Haemorrhage-non-SAE, NR, Severe | 0 | 1
  Gastrooesophageal Reflux Disease-non-SAE, NR, Mild | 1 | 2
  Gastrooesophageal Reflux Disease-non-SAE, NR, Mod | 1 | 0
  Genital Herpes-non-SAE, NR, Mild | 1 | 0
  Genital Swelling-non-SAE, Rboth, Mod | 0 | 1
  Goitre-non-SAE, NR, Mild | 1 | 0
  Gout-non-SAE, NR, Mild | 0 | 1
  Grand Mal Convulsion-non-SAE, NR, Severe | 1 | 0
  Grand Mal Convulsion-SAE, NR, Severe | 0 | 1
  Gravitational Oedema-non-SAE, Rboth, Mod | 0 | 1
  Groin Pain-non-SAE, NR, Mild | 0 | 1
  Groin Pain-non-SAE, RIGIV, Mild | 0 | 1
  Groin Pain-non-SAE, RrHu, Mod | 0 | 1
  Haematoma-non-SAE, NR, Mild | 1 | 1
  Haematoma-non-SAE, NR, Mod | 0 | 1
  Haematuria-non-SAE, NR, Mild | 0 | 1
  Haemoglobin Abnormal-non-SAE, NR, Mild | 0 | 1
  Haemorrhoids-non-SAE, NR, Mild | 0 | 2
  Hand Fracture-non-SAE, NR, Mod | 0 | 1
  Headache-non-SAE, NR, Mild | 13 | 16
  Headache-non-SAE, NR, Mod | 1 | 3
  Headache-non-SAE, NR, Severe | 1 | 0
  Headache-non-SAE, RIGIV, Mild | 25 | 14
  Headache-non-SAE, RIGIV, Mod | 12 | 5
  Headache-non-SAE, RIGIV, Severe | 1 | 0
  Headache-non-SAE, Rboth, Mild | 0 | 9
  Headache-non-SAE, Rboth, Mod | 0 | 8
  Headache-SAE, NR, Severe | 0 | 1
  Hearing Impaired-non-SAE, NR, Mild | 0 | 1
  Heart Rate Increased-non-SAE, RIGIV, Mild | 4 | 0
  Heat Rash-non-SAE, NR, Mild | 0 | 1
  Heat Stroke-non-SAE, NR, Mod | 0 | 1
  Herpes Simplex Ophthalmic-non-SAE, NR, Mod | 0 | 1
  Herpes Zoster-non-SAE, NR, Mod | 0 | 1
  Hiatus Hernia-non-SAE, NR, Mod | 0 | 1
  Hot Flush-non-SAE, RIGIV, Mild | 1 | 0
  Hyperaesthesia-non-SAE, NR, Mild | 0 | 1
  Hypercholesterolaemia-non-SAE, NR, Mod | 0 | 1
  Hyperkeratosis-non-SAE, NR, Mild | 0 | 1
  Hypertension-non-SAE, NR, Mod | 0 | 4
  Hypertension-non-SAE, RIGIV, Mild | 0 | 2
  Hypertension-non-SAE, RIGIV, Mod | 0 | 1
  Hypertonia-non-SAE, NR, Mild | 0 | 1
  Hypothyroidism-non-SAE, NR, Mild | 0 | 1
  Idiopathic Urticaria-non-SAE, NR, Mod | 1 | 0
  Increased Upper Airway Secretion-non-SAE, NR, Mild | 2 | 0
  Infected Bites-non-SAE, NR, Mild | 0 | 2
  Infected Bites-non-SAE, NR, Mod | 1 | 1
  Infection-non-SAE, NR, Mod | 0 | 2
  Influenza-non-SAE, NR, Mild | 1 | 2
  Influenza-non-SAE, NR, Mod | 4 | 3
  Influenza Like Illness-non-SAE, NR, Mild | 0 | 1
  Infusion Related Reaction-non-SAE, RIGIV, Mild | 0 | 1
  Infusion Related Reaction-non-SAE, RIGIV, Mod | 1 | 0
  Infusion Related Reaction-non-SAE, Rboth, Mild | 0 | 1
  Infusion Related Reaction-non-SAE, Rboth, Mod | 0 | 1
  Infusion Site Discomfort-non-SAE, RIGIV, Mild | 0 | 6
  Infusion Site Discomfort-non-SAE, RrHu, Mod | 0 | 1
  Infusion Site Discomfort-non-SAE, Rboth, Mild | 0 | 15
  Infusion Site Discomfort-non-SAE, Rboth, Mod | 0 | 8
  Infusion Site Erythema-non-SAE, RIGIV, Mild | 0 | 1
  Infusion Site Erythema-non-SAE, RrHu, Mild | 0 | 2
  Infusion Site Erythema-non-SAE, Rboth, Mild | 0 | 20
  Infusion Site Erythema-non-SAE, Rboth, Mod | 0 | 5
  Infusion Site Extravasation-non-SAE, NR, Mild | 2 | 0
  Infusion Site Haematoma-non-SAE, RIGIV, Mild | 0 | 1
  Infusion Site Haemorrhage-non-SAE, Rboth, Mild | 0 | 1
  Infusion Site Hypersensitivity-non-SAE, NR, Severe | 0 | 1
  Infusion Site Hypersensitivity-non-SAE, Rboth, Mod | 0 | 1
  Infusion Site Mass-non-SAE, RIGIV, Mild | 0 | 1
  Infusion Site Mass-non-SAE, Rboth, Mild | 0 | 2
  Infusion Site Oedema-non-SAE, Rboth, Mild | 0 | 4
  Infusion Site Oedema-non-SAE, Rboth, Mod | 0 | 5
  Infusion Site Pain-non-SAE, NR, Mild | 0 | 2
  Infusion Site Pain-non-SAE, RIGIV, Mild | 1 | 12
  Infusion Site Pain-non-SAE, RIGIV, Mod | 0 | 6
  Infusion Site Pain-non-SAE, RrHu, Mild | 0 | 35
  Infusion Site Pain-non-SAE, RrHu, Mod | 0 | 1
  Infusion Site Pain-non-SAE, Rboth, Mild | 0 | 19
  Infusion Site Pain-non-SAE, Rboth, Mod | 0 | 16
  Infusion Site Pain-non-SAE, Rboth, Severe | 0 | 1
  Infusion Site Pruritus-non-SAE, RIGIV, Mild | 0 | 2
  Infusion Site Pruritus-non-SAE, RrHu, Mild | 0 | 5
  Infusion Site Pruritus-non-SAE, Rboth, Mild | 0 | 6
  Infusion Site Pruritus-non-SAE, Rboth, Mod | 0 | 4
  Infusion Site Reaction-non-SAE, Rboth, Mild | 0 | 1
  Infusion Site Reaction-non-SAE, Rboth, Mod | 0 | 2
  Infusion Site Swelling-non-SAE, RIGIV, Mild | 0 | 2
  Infusion Site Swelling-non-SAE, Rboth, Mild | 0 | 3
  Infusion Site Swelling-non-SAE, Rboth, Mod | 0 | 4
  Infusion Site Swelling-non-SAE, Rboth, Severe | 0 | 1
  Infusion Site Warmth-non-SAE, Rboth, Mild | 0 | 2
  Ingrowing Nail-non-SAE, NR, Mod | 0 | 1
  Injection Site Erythema-non-SAE, RIGIV, Mild | 0 | 1
  Injury-non-SAE, NR, Mild | 1 | 0
  Insomnia-non-SAE, NR, Mild | 1 | 0
  Intervertebral Disc Protrusion-non-SAE, NR, Mod | 1 | 0
  Irritable Bowel Syndrome-non-SAE, NR, Mild | 0 | 1
  Irritable Bowel Syndrome-non-SAE, NR, Mod | 0 | 2
  Joint Effusion-non-SAE, NR, Mild | 0 | 1
  Joint Effusion-non-SAE, NR, Mod | 0 | 1
  Joint Injury-non-SAE, NR, Mod | 1 | 1
  Joint Range of Motion Decreased-non-SAE, NR, Mod | 0 | 2
  Joint Sprain-non-SAE, NR, Mild | 0 | 1
  Joint Sprain-non-SAE, NR, Mod | 0 | 2
  Joint Swelling-non-SAE, NR, Mild | 0 | 1
  Jugular Vein Distension-non-SAE, NR, Mild | 0 | 1
  Lethargy-non-SAE, NR, Mild | 0 | 1
  Lethargy-non-SAE, RIGIV, Mod | 1 | 0
  Ligament Injury-non-SAE, NR, Mod | 0 | 1
  Ligament Sprain-non-SAE, NR, Mod | 0 | 1
  Limb Injury-non-SAE, NR, Mild | 1 | 0
  Lip Injury-non-SAE, NR, Mild | 0 | 1
  Lip Ulceration-non-SAE, NR, Mild | 0 | 1
  Local Swelling-non-SAE, RIGIV, Mild | 0 | 3
  Local Swelling-non-SAE, Rboth, Mild | 0 | 3
  Localised Infection-non-SAE, NR, Mild | 0 | 1
  Localised Oedema-non-SAE, RIGIV, Mild | 0 | 1
  Localised Oedema-non-SAE, Rboth, Mod | 0 | 1
  Lung Infection-non-SAE, NR, Mod | 1 | 0
  Lung Infection-non-SAE, NR, Severe | 1 | 0
  Lymph Gland Infection-non-SAE, NR, Mod | 1 | 0
  Lymph Node Pain-non-SAE, NR, Mild | 1 | 0
  Lymph Node Pain-non-SAE, NR, Mod | 0 | 1
  Lymph Node Palpable-non-SAE, NR, Mild | 1 | 0
  Lymphadenitis-non-SAE, NR, Mod | 1 | 0
  Lymphadenopathy-non-SAE, NR, Mild | 2 | 8
  Lymphangitis-non-SAE, NR, Mod | 0 | 1
  Lymphocyte Count Decreased-non-SAE, RIGIV, Mild | 0 | 1
  Lymphoedema-non-SAE, NR, Severe | 1 | 0
  Malaise-non-SAE, NR, Mild | 0 | 2
  Malaise-non-SAE, NR, Mod | 0 | 1
  Malaise-non-SAE, RIGIV, Mod | 1 | 0
  Malaise-non-SAE, RrHu, Mild | 0 | 1
  Malaise-non-SAE, RrHu, Mod | 0 | 1
  Memory Impairment-non-SAE, NR, Mod | 0 | 1
  Migraine-non-SAE, NR, Mild | 1 | 1
  Migraine-non-SAE, NR, Mod | 0 | 2
  Migraine-non-SAE, NR, Severe | 1 | 0
  Migraine-non-SAE, RIGIV, Mild | 1 | 1
  Migraine-non-SAE, RIGIV, Mod | 1 | 4
  Migraine-non-SAE, RIGIV, Severe | 0 | 1
  Migraine-non-SAE, Rboth, Mod | 0 | 1
  Molluscum Contagiosum-non-SAE, NR, Mild | 2 | 0
  Mouth Ulceration-non-SAE, NR, Mild | 1 | 0
  Multiple Sclerosis Relapse-non-SAE, NR, Mod | 0 | 1
  Muscle Fatigue-non-SAE, NR, Mild | 0 | 1
  Muscle Injury-non-SAE, NR, Mild | 0 | 2
  Muscle Spasms-non-SAE, NR, Mild | 0 | 1
  Muscle Spasms-non-SAE, RIGIV, Mild | 1 | 0
  Muscle Strain-non-SAE, NR, Mild | 1 | 1
  Muscle Strain-non-SAE, NR, Mod | 0 | 1
  Muscular Weakness-non-SAE, NR, Mild | 1 | 0
  Musculoskeletal Chest Pain-non-SAE, NR, Mild | 0 | 1
  Musculoskeletal Chest Pain-non-SAE, RIGIV, Mild | 0 | 1
  Musculoskeletal Pain-non-SAE, NR, Mild | 2 | 0
  Musculoskeletal Pain-non-SAE, NR, Mod | 1 | 1
  Musculoskeletal Stiffness-non-SAE, NR, Mild | 1 | 1
  Myalgia-non-SAE, NR, Mild | 3 | 5
  Myalgia-non-SAE, NR, Mod | 1 | 4
  Myalgia-non-SAE, NR, Severe | 0 | 1
  Myalgia-non-SAE, RIGIV, Mild | 0 | 6
  Myalgia-non-SAE, RIGIV, Mod | 1 | 1
  Myalgia-non-SAE, Rboth, Mild | 0 | 3

53. Secondary Outcome: Number of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to Study Drug, and Severity (N-Z)
Description: Categories presented as Preferred term-Seriousness, Relatedness, Severity. The following codes are to be used: Seriousness: non-SAE-non-serious AE; SAE-serious AE Relationship: NR-not related to immune globulin (IGIV), 10% and recombinant human hyaluronidase (rHuPH20); RIGIV-related to IGIV, 10%; RrHu-related to rHuPH20; Rboth-related to both IGIV, 10% and rHuPH20 Severity: Mild; Mod (Moderate); Severe Preferred terms abbreviated: Resp.-Respiratory WBC - White blood cells
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number of AEs
  Nasal Congestion-non-SAE, NR, Mild | 4 | 3
  Nasal Congestion-non-SAE, NR, Mod | 0 | 2
  Nasal Congestion-non-SAE, RIGIV, Mild | 0 | 3
  Nasal Discomfort-non-SAE, NR, Mild | 0 | 1
  Nasal Mucosal Discolouration-non-SAE, NR, Mild | 0 | 1
  Nasal Turbinate Hypertrophy-non-SAE, NR, Mild | 0 | 1
  Nasopharyngitis-non-SAE, NR, Mild | 4 | 8
  Nausea-non-SAE, NR, Mild | 3 | 17
  Nausea-non-SAE, NR, Mod | 2 | 3
  Nausea-non-SAE, RIGIV, Mild | 7 | 1
  Nausea-non-SAE, RIGIV, Mod | 1 | 0
  Nausea-non-SAE, Rboth, Mild | 0 | 4
  Neck Pain-non-SAE, NR, Mild | 1 | 1
  Night Sweats-non-SAE, NR, Mild | 1 | 0
  Night Sweats-non-SAE, NR, Mod | 0 | 1
  Nodule-non-SAE, Rboth, Mild | 0 | 2
  Oedema-non-SAE, RIGIV, Mild | 0 | 1
  Oedema Genital-non-SAE, Rboth, Severe | 0 | 1
  Oedema Peripheral-non-SAE, NR, Mild | 0 | 1
  Oedema Peripheral-non-SAE, NR, Mod | 0 | 1
  Oedema Peripheral-non-SAE, Rboth, Mod | 0 | 2
  Oesophagitis-non-SAE, NR, Mild | 0 | 1
  Onychomycosis-non-SAE, NR, Mild | 0 | 1
  Oral Candidiasis-non-SAE, NR, Mod | 0 | 1
  Oral Fungal Infection-non-SAE, NR, Mild | 0 | 1
  Oral Herpes-non-SAE, NR, Mild | 1 | 2
  Oral Herpes-non-SAE, NR, Mod | 0 | 1
  Oral Pain-non-SAE, NR, Mild | 0 | 1
  Oral Pain-non-SAE, RrHu, Severe | 0 | 1
  Oropharyngeal Pain-non-SAE, NR, Mild | 1 | 4
  Oropharyngeal Pain-non-SAE, NR, Mod | 2 | 1
  Osteoarthritis-non-SAE, NR, Mod | 0 | 1
  Osteopenia-non-SAE, NR, Mild | 0 | 1
  Osteopenia-non-SAE, NR, Mod | 0 | 1
  Osteoporosis-non-SAE, NR, Mild | 0 | 1
  Otitis Externa-non-SAE, NR, Mild | 0 | 1
  Otitis Externa-non-SAE, NR, Mod | 0 | 1
  Otitis Media-non-SAE, NR, Mod | 1 | 1
  Pain-non-SAE, NR, Mild | 1 | 5
  Pain-non-SAE, NR, Mod | 1 | 1
  Pain-non-SAE, RIGIV, Mild | 0 | 1
  Pain-non-SAE, RIGIV, Mod | 2 | 1
  Pain-non-SAE, Rboth, Mild | 0 | 1
  Pain-non-SAE, Rboth, Mod | 0 | 1
  Pain in Extremity-non-SAE, NR, Mild | 2 | 1
  Pain in Extremity-non-SAE, NR, Mod | 1 | 2
  Pain in Extremity-non-SAE, RIGIV, Mod | 2 | 0
  Pain in Extremity-non-SAE, RIGIV, Severe | 1 | 0
  Pain in Extremity-non-SAE, Rboth, Mild | 0 | 3
  Pain in Extremity-non-SAE, Rboth, Mod | 0 | 2
  Palpitations-non-SAE, NR, Mild | 1 | 1
  Papule-non-SAE, NR, Mild | 0 | 1
  Peptic Ulcer Haemorrhage-SAE, NR, Severe | 1 | 0
  Periorbital Haematoma-non-SAE, NR, Mild | 0 | 1
  Peripheral Nerve Injury-non-SAE, NR, Mild | 0 | 1
  Pertussis-non-SAE, NR, Mod | 0 | 1
  Petit Mal Epilepsy-SAE, NR, Severe | 0 | 1
  Pharyngeal Erythema-non-SAE, NR, Mild | 1 | 3
  Pharyngitis-non-SAE, NR, Mild | 1 | 4
  Pharyngitis-non-SAE, NR, Mod | 1 | 0
  Pharyngitis Streptococcal-non-SAE, NR, Mod | 0 | 4
  Pneumonia-non-SAE, NR, Mild | 0 | 1
  Pneumonia-non-SAE, NR, Mod | 0 | 1
  Pneumonia Bacterial-non-SAE, NR, Mod | 0 | 1
  Post Procedural Infection-non-SAE, NR, Mild | 1 | 2
  Post Procedural Infection-non-SAE, NR, Mod | 0 | 5
  Postictal Paralysis-non-SAE, NR, Mod | 0 | 1
  Postoperative Wound Infection-non-SAE, NR, Mod | 0 | 1
  Procedural Pain-non-SAE, NR, Mild | 0 | 2
  Procedural Pain-non-SAE, NR, Mod | 0 | 1
  Productive Cough-non-SAE, NR, Mild | 1 | 1
  Pruritus-non-SAE, NR, Mild | 1 | 0
  Pruritus-non-SAE, RIGIV, Mild | 1 | 0
  Pruritus-non-SAE, Rboth, Mild | 0 | 1
  Pruritus-non-SAE, Rboth, Mod | 0 | 1
  Pruritus Generalized-non-SAE, NR, Mild | 1 | 0
  Pseudomonas Infection-non-SAE, NR, Mod | 0 | 1
  Psoriasis-non-SAE, NR, Mod | 0 | 1
  Pyrexia-non-SAE, NR, Mild | 3 | 11
  Pyrexia-non-SAE, NR, Mod | 2 | 1
  Pyrexia-non-SAE, RIGIV, Mild | 4 | 6
  Pyrexia-non-SAE, RIGIV, Mod | 2 | 2
  Pyrexia-non-SAE, Rboth, Mild | 0 | 2
  Rales-non-SAE, NR, Mild | 0 | 1
  Rales-non-SAE, NR, Mod | 0 | 1
  Rash-non-SAE, NR, Mild | 2 | 5
  Rash-non-SAE, NR, Mod | 0 | 1
  Rash Erythematous-non-SAE, NR, Mild | 0 | 1
  Rash Macro-Papular-non-SAE, Rboth, Mild | 0 | 1
  Rash Pustular-non-SAE, NR, Mild | 0 | 1
  Rash Pustular-non-SAE, NR, Mod | 1 | 0
  Rash Papular-non-SAE, NR, Mild | 0 | 1
  Respiratory Failure-SAE, NR, Severe | 0 | 1
  Respiratory Rate Increased-non-SAE, NR, Mild | 0 | 1
  Respiratory Tract Congestion-non-SAE, NR, Mild | 0 | 1
  Respiratory Tract Infection-non-SAE, NR, Mild | 1 | 1
  Respiratory Tract Infection-non-SAE, NR, Mod | 1 | 3
  Respiratory Tract Infection Viral-non-SAE, NR, Mod | 1 | 0
  Rhinitis Allergic-non-SAE, NR, Mild | 1 | 3
  Rhinitis Allergic-non-SAE, NR, Mod | 3 | 1
  Rhinitis Allergic-non-SAE, RIGIV, Mod | 1 | 0
  Rhinorrhoea-non-SAE, NR, Mild | 1 | 1
  Road Traffic Accident-non-SAE, NR, Mod | 0 | 2
  Scleritis-non-SAE, NR, Mild | 1 | 1
  Scleritis-non-SAE, NR, Mod | 0 | 1
  Scratch-non-SAE, NR, Mild | 1 | 0
  Seborrhoeic Dermatitis-non-SAE, NR, Mild | 0 | 1
  Sicca Syndrome-non-SAE, NR, Mod | 0 | 1
  Sinus Congestion-non-SAE, NR, Mild | 1 | 0
  Sinus Headache-non-SAE, NR, Mild | 1 | 0
  Sinusitis-non-SAE, NR, Mild | 6 | 25
  Sinusitis-non-SAE, NR, Mod | 13 | 26
  Sinusitis-non-SAE, NR, Severe | 0 | 1
  Sinusitis-non-SAE, RIGIV, Mod | 0 | 1
  Skeletal Injury-non-SAE, NR, Mild | 0 | 1
  Skeletal Injury-non-SAE, NR, Mod | 0 | 1
  Skin Hyperpigmentation-non-SAE, Rboth, Mild | 0 | 1
  Skin Laceration-non-SAE, NR, Mild | 0 | 1
  Skin Laceration-non-SAE, NR, Mod | 0 | 1
  Skin Lesion-non-SAE, NR, Mild | 2 | 1
  Skin Lesion-non-SAE, NR, Mod | 1 | 0
  Skin Lesion-non-SAE, RIGIV, Mild | 0 | 2
  Skin Papilloma-non-SAE, NR, Mod | 1 | 0
  Spinal Osteoarthritis-non-SAE, NR, Mild | 0 | 2
  Squamous Cell Carcinoma-non-SAE, NR, Mod | 1 | 1
  Status Epilepticus-SAE, NR, Severe | 0 | 1
  Suicidal Ideation-non-SAE, NR, Mild | 1 | 0
  Sunburn-non-SAE, NR, Mild | 0 | 1
  Swelling-non-SAE, Rboth, Mild | 0 | 1
  Swelling-non-SAE, Rboth, Mod | 0 | 3
  Syncope-non-SAE, NR, Mild | 0 | 1
  Tachycardia-non-SAE, NR, Mild | 0 | 3
  Tachycardia-non-SAE, NR, Mod | 0 | 1
  Therapy Cessation-non-SAE, NR, Severe | 0 | 1
  Thrombosis-non-SAE, NR, Severe | 0 | 1
  Thrombosis-SAE, NR, Mod | 0 | 1
  Tinea Infection-non-SAE, NR, Mild | 2 | 0
  Tongue Coated-non-SAE, NR, Mild | 0 | 1
  Tonsillar Hypertrophy-non-SAE, NR, Mod | 0 | 1
  Tonsillar Hypertrophy-SAE, NR, Mild | 0 | 1
  Tooth Abscess-non-SAE, NR, Mild | 1 | 0
  Tooth Abscess-non-SAE, NR, Mod | 0 | 1
  Tooth Impacted-non-SAE, NR, Mod | 0 | 1
  Tooth Infection-non-SAE, NR, Mod | 0 | 1
  Toothache-non-SAE, NR, Mod | 0 | 1
  Tongue Injury-non-SAE, NR, Mild | 0 | 1
  Tremor-non-SAE, NR, Mild | 0 | 1
  Tricuspid Valve Incompetence-non-SAE, NR, Mild | 0 | 1
  Tympanic Membrane Disorder-non-SAE, NR, Mild | 1 | 0
  Tympanic Membrane Hyperaemia-non-SAE, NR, Mild | 0 | 2
  Upper Airway Cough Syndrome-non-SAE, NR, Mild | 0 | 1
  Upper Resp. Tract Infection-non-SAE, NR, Mild | 7 | 34
  Upper Resp. Tract Infection-non-SAE, NR, Mod | 2 | 10
  Urinary Tract Infection-non-SAE, NR, Mild | 1 | 2
  Urinary Tract Infection-non-SAE, NR, Mod | 5 | 4
  Urine Analysis Abnormal-non-SAE, NR, Mild | 0 | 1
  Urticaria-non-SAE, NR, Mild | 0 | 5
  Urticaria-non-SAE, NR, Mod | 0 | 1
  Urticaria-non-SAE, RIGIV, Mild | 1 | 0
  Uterine Polyp-non-SAE, NR, Mod | 0 | 1
  Vaginal Haemorrhage-non-SAE, NR, Mod | 0 | 1
  Vascular Access Complication-non-SAE, NR, Mild | 1 | 0
  Vertigo-non-SAE, NR, Mod | 0 | 1
  Viral Diarrhoea-non-SAE, NR, Mild | 0 | 1
  Viral Infection-non-SAE, NR, Mild | 3 | 7
  Viral Infection-non-SAE, NR, Mod | 3 | 3
  Viral Infection-SAE, NR, Mild | 1 | 0
  Viral Upper Resp. Tract Infection-non-SAE, NR Mild | 1 | 8
  Viral Upper Resp. Tract Infection-non-SAE, NR, Mod | 1 | 1
  Vision Blurred-non-SAE, NR, Mild | 0 | 1
  Vitamin D Deficiency-non-SAE, NR, Mild | 1 | 0
  Vitamin D Deficiency-non-SAE, NR, Mod | 0 | 2
  Vomiting-non-SAE, NR, Mild | 5 | 7
  Vomiting-non-SAE, NR, Mod | 0 | 3
  Vomiting-non-SAE, RIGIV, Mild | 4 | 3
  Vomiting-non-SAE, RIGIV, Mod | 1 | 4
  Vomiting-non-SAE, RIGIV, Severe | 1 | 0
  Vomiting-non-SAE, Rboth, Mod | 0 | 1
  Vulvovaginal Pruritus-non-SAE, RIGIV, Mild | 0 | 1
  Weight Decreased-non-SAE, RrHu, Mild | 0 | 1
  Weight Decreased-non-SAE, RrHu, Mod | 0 | 1
  Wheezing-non-SAE, NR, Mod | 0 | 1
  WBC Count Decreased-non-SAE, RIGIV, Mild | 0 | 1
  White Blood Cells Urine Positive-non-SAE, NR, Mild | 0 | 1
  WBC Urine Positive-non-SAE, RIGIV Mild | 1 | 0

54. Secondary Outcome: Rate of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to Study Drug, and Severity Per Infusion (A-F)
Description: as for outcome 51
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Number of AEs per infusion
  Abdominal Discomfort-non-SAE, NR, Mod | 0 | 0.001
  Abdominal Distension-non-SAE, Rboth, Mild | 0 | 0.001
  Abdominal Hernia-non-SAE, NR, Mild | 0 | 0.001
  Abdominal Pain-non-SAE, NR, Mild | 0.003 | 0.002
  Abdominal Pain-non-SAE, NR, Mod | 0 | 0.001
  Abdominal Pain-non-SAE, Rboth, Mild | 0 | 0.003
  Abdominal Pain-non-SAE, Rboth, Mod | 0 | 0.001
  Abdominal Pain Lower-non-SAE, NR, Mild | 0 | 0.001
  Abdominal Pain Upper-non-SAE, NR, Mild | 0.003 | 0.004
  Abdominal Pain Upper-non-SAE, NR, Mod | 0.003 | 0
  Abdominal Pain Upper-non-SAE, RIGIV, Mild | 0 | 0.001
  Abdominal Pain Upper-non-SAE, RIGIV, Mod | 0.003 | 0
  Abdominal Pain Upper-non-SAE, Rboth, Mild | 0 | 0.002
  Abdominal Tenderness-non-SAE, NR, Mod | 0.003 | 0
  Abdominal Tenderness-non-SAE, RIGIV, Mild | 0 | 0.001
  Abdominal Tenderness-non-SAE, RIGIV, Mod | 0 | 0.002
  Acarodermatitis-non-SAE, NR, Mild | 0 | 0.001
  Acne-non-SAE, NR, Mild | 0.003 | 0.001
  Acute Sinusitis-non-SAE, NR, Mild | 0.003 | 0
  Acute Sinusitis-non-SAE, NR, Mod | 0 | 0.004
  Adenoidal Hypertrophy-non-SAE, NR, Mod | 0 | 0.001
  Adnexa Uteri Cyst-non-SAE, NR, Mild | 0.003 | 0
  Adrenocortical Insufficiency Acute-SAE, NR, Mod | 0 | 0.001
  Allergic Respiratory Symptom-non-SAE, NR, Mild | 0 | 0.001
  Allergic Sinusitis-non-SAE, NR, Mild | 0.003 | 0
  Alopecia-non-SAE, NR, Mild | 0.003 | 0
  Animal Bite-non-SAE, NR, Mod | 0.003 | 0
  Antibody Test Positive-non-SAE, Rboth, Mod | 0 | 0.001
  Anxiety-non-SAE, NR, Mild | 0 | 0.001
  Anxiety-non-SAE, NR, Mod | 0.003 | 0
  Aphthous Stomatitis-non-SAE, NR, Mild | 0.005 | 0.001
  Aphthous Stomatitis-non-SAE, NR, Mod | 0 | 0.001
  Arteriosclerosis Coronary Artery-non-SAE, NR, Mild | 0 | 0.001
  Arthralgia-non-SAE, NR, Mild | 0 | 0.004
  Arthralgia-non-SAE, NR, Mod | 0.003 | 0.005
  Arthralgia-non-SAE, RIGIV, Mild | 0 | 0.001
  Arthralgia-non-SAE, RIGIV, Mod | 0 | 0.002
  Arthritis-non-SAE, NR, Mod | 0.003 | 0.001
  Arthropathy-non-SAE, NR, Mod | 0.003 | 0
  Arthropod Bite-non-SAE, NR, Mild | 0.005 | 0.002
  Arthropod Sting-non-SAE, NR, Mild | 0 | 0.001
  Arthropod Sting-non-SAE, NR, Mod | 0.003 | 0
  Aspiration-non-SAE, NR, Mild | 0 | 0.001
  Asthenia-non-SAE, NR, Mild | 0 | 0.003
  Asthenia-non-SAE, NR, Mod | 0.003 | 0
  Asthenia-non-SAE, RIGIV, Mild | 0 | 0.001
  Asthma-non-SAE, NR, Mild | 0 | 0.004
  Asthma-non-SAE, NR, Mod | 0.022 | 0.019
  Asthma-non-SAE, NR, Severe | 0 | 0.001
  ADHD-non-SAE, NR, Mod | 0 | 0.001
  Back Injury-non-SAE, NR, Mod | 0.003 | 0
  Back Injury-SAE, NR, Severe | 0 | 0.001
  Back Pain-non-SAE, NR, Mild | 0.003 | 0.002
  Back Pain-non-SAE, NR, Mod | 0.003 | 0.004
  Bacterial Prostatitis-non-SAE, NR, Mild | 0 | 0.001
  Blepharitis-non-SAE, NR, Mod | 0.003 | 0
  Blister-non-SAE, NR, Mild | 0 | 0.001
  Blood Pressure Decreased-non-SAE, NR, Mild | 0 | 0.001
  Blood Pressure Decreased-non-SAE, Rboth, Mild | 0 | 0.001
  Blood Pressure Increased-non-SAE, NR, Mod | 0 | 0.001
  Blood Pressure Increased-non-SAE, RIGIV, Mild | 0 | 0.001
  Blood Pressure Increased-non-SAE, RIGIV, Mod | 0 | 0.001
  Blood Pressure Increased-non-SAE, RrHu, Mild | 0 | 0.001
  BP Systolic Increased-non-SAE, RIGIV, Mild | 0.003 | 0
  Blood Urea Increased-non-SAE, NR, Mild | 0 | 0.001
  Body Fat Disorder-non-SAE, NR, Mild | 0 | 0.001
  Body Tinea-non-SAE, NR, Mild | 0.003 | 0
  Body Tinea-non-SAE, NR, Mod | 0 | 0.001
  Bone Pain-non-SAE, NR, Mild | 0 | 0.001
  Breast Pain-non-SAE, NR, Mild | 0.003 | 0
  Bronchal Hyperreactivity-non-SAE, NR, Mild | 0 | 0.001
  Bronchitis-non-SAE, NR, Mild | 0.011 | 0.002
  Bronchitis-non-SAE, NR, Mod | 0.005 | 0.007
  Bronchitis-SAE, NR, Mod | 0.003 | 0
  Bronchospasm-non-SAE, NR, Mod | 0 | 0.001
  Burn Infection-non-SAE, NR, Mild | 0 | 0.001
  Burning Sensation-non-SAE, RIGIV, Mild | 0 | 0.001
  Burning Sensation-non-SAE, RIGIV, Mod | 0 | 0.001
  Burning Sensation-non-SAE, RrHu, Mild | 0 | 0.001
  Bursitis-non-SAE, NR, Mild | 0.003 | 0
  Bursitis-non-SAE, NR, Mod | 0 | 0.001
  Candidiasis-non-SAE, NR, Mild | 0.003 | 0
  Candidiasis-non-SAE, NR, Mod | 0.003 | 0.001
  Cardiac Murmur-non-SAE, NR, Mild | 0 | 0.001
  Cellulitis-non-SAE, NR, Mild | 0 | 0.001
  Cellulitis-non-SAE, NR, Mod | 0 | 0.003
  Cellulitis-non-SAE, Rboth, Mod | 0 | 0.001
  Cerumen Impaction-non-SAE, NR, Mild | 0 | 0.002
  Cervical Dysplasia-SAE, NR, Mild | 0.003 | 0.001
  Cheilitis-non-SAE, NR, Mild | 0.005 | 0
  Chest Pain-non-SAE, NR, Mild | 0 | 0.002
  Chills-non-SAE, NR, Mild | 0 | 0.003
  Chills-non-SAE, RIGIV, Mild | 0.016 | 0.001
  Chills-non-SAE, RIGIV, Mod | 0.008 | 0
  Chills-non-SAE, Rboth, Mild | 0 | 0.001
  COPD-non-SAE, NR, Mod | 0 | 0.002
  COPD-non-SAE, NR, Severe | 0.003 | 0
  Chronic Sinusitis-non-SAE, NR, Mild | 0 | 0.004
  Chronic Sinusitis-non-SAE, NR, Mod | 0.003 | 0.001
  Concussion-non-SAE, NR, Mod | 0.003 | 0
  Confusional State-non-SAE, NR, Mod | 0 | 0.001
  Confusional State-non-SAE, RIGIV, Mild | 0.003 | 0
  Conjunctivitis-non-SAE, NR, Mild | 0.003 | 0.002
  Conjunctivitis Allergic-non-SAE, NR, Mild | 0.003 | 0
  Conjunctivitis Allergic-non-SAE, NR, Mod | 0.003 | 0
  Conjunctivitis Bacterial-non-SAE, NR, Mild | 0.003 | 0.001
  Conjunctivitis Bacterial-non-SAE, NR, Mod | 0 | 0.001
  Conjunctivitis Bacterial-non-SAE, NR, Severe | 0 | 0.001
  Constipation-non-SAE, NR, Mild | 0 | 0.003
  Contusion-non-SAE, NR, Mild | 0.003 | 0.004
  Contusion-non-SAE, NR, Mod | 0.003 | 0
  Contusion-non-SAE, RIGIV, Mod | 0 | 0.001
  Coombs Test Positive-non-SAE, RIGIV, Mild | 0 | 0.001
  Costochondritis-non-SAE, NR, Mod | 0 | 0.001
  Cough-non-SAE, NR, Mild | 0.008 | 0.005
  Cough-non-SAE, NR, Mod | 0 | 0.002
  Cough-non-SAE, RIGIV, Mild | 0.003 | 0
  Cushingoid-non-SAE, NR, Mild | 0 | 0.001
  Cystitis-non-SAE, NR, Mild | 0 | 0.001
  Deafness Neurosensory-non-SAE, NR, Mild | 0.003 | 0
  Decreased Appetite-non-SAE, NR, Mild | 0.003 | 0.001
  Decreased Appetite-non-SAE, RrHu, Mild | 0 | 0.001
  Decreased Appetite-non-SAE, Rboth, Mild | 0 | 0.002
  Dehydration-non-SAE, NR, Mod | 0 | 0.002
  Dental Caries-non-SAE, NR, Mild | 0 | 0.002
  Dental Caries-non-SAE, NR, Mod | 0 | 0.003
  Depressed Mood-non-SAE, NR, Mild | 0 | 0.001
  Depression-non-SAE, NR, Severe | 0 | 0.001
  Dermal Cyst-non-SAE, NR, Mild | 0 | 0.001
  Dermatitis-non-SAE, NR, Mild | 0 | 0.002
  Dermatitis-non-SAE, NR, Mod | 0.003 | 0
  Dermatitis Acneiform-non-SAE, NR, Mod | 0.003 | 0
  Dermatitis Contact-non-SAE, NR, Mild | 0 | 0.002
  Dermatitis Contact-non-SAE, NR, Mod | 0.005 | 0.002
  Dermatitis Infected-non-SAE, NR, Mild | 0 | 0.002
  Dermatitis Infected-non-SAE, NR, Mod | 0 | 0.001
  Dermatitis Infected-non-SAE, NR, Severe | 0 | 0.001
  Device Failure-non-SAE, NR, Mild | 0.005 | 0.001
  Device Failure-non-SAE, NR, Mod | 0 | 0.002
  Diarrhoea-non-SAE, NR, Mild | 0.008 | 0.005
  Diarrhoea-non-SAE, NR, Mod | 0.005 | 0.004
  Diarrhoea-non-SAE, RIGIV, Mild | 0.003 | 0.001
  Diarrhoea-non-SAE, RIGIV, Mod | 0.003 | 0
  Diarrhoea Haemorrhagic-non-SAE, NR, Mild | 0.003 | 0
  Diarrhoea Infectious-non-SAE, NR, Mild | 0 | 0.001
  Diastolic Dysfunction-non-SAE, NR, Mild | 0 | 0.001
  Disaccharide Metabolism Disorder-non-SAE, NR, Mild | 0 | 0.001
  Disturbance in Attention-non-SAE, NR, Mild | 0 | 0.002
  Diverticulitis-non-SAE, NR, Mod | 0.003 | 0
  Dizziness-non-SAE, NR, Mild | 0.005 | 0.006
  Dizziness-non-SAE, NR, Mod | 0 | 0.002
  Dizziness-non-SAE, RIGIV, Mild | 0 | 0.003
  Dizziness-non-SAE, RIGIV, Mod | 0.003 | 0
  Drug Eruption-non-SAE, NR, Mod | 0.003 | 0
  Dry Eye-non-SAE, NR, Mod | 0 | 0.001
  Dry Mouth-non-SAE, NR, Mild | 0 | 0.001
  Dry Skin-non-SAE, NR, Mild | 0 | 0.003
  Dysmenorrhoea-non-SAE, NR, Mild | 0 | 0.001
  Dyspepsia-non-SAE, NR, Mild | 0 | 0.002
  Dyspepsia-non-SAE, NR, Mod | 0 | 0.001
  Dyspepsia-non-SAE, RIGIV, Mild | 0.003 | 0
  Dysphagia-non-SAE, NR, Mild | 0 | 0.001
  Dysphagia-non-SAE, NR, Mod | 0 | 0.001
  Dyspnoea-non-SAE, NR, Mild | 0.003 | 0
  Dyspnoea-non-SAE, NR, Mod | 0.003 | 0
  Dyspnoea-non-SAE, RIGIV, Mild | 0.003 | 0
  Dysuria-non-SAE, NR, Mild | 0 | 0.002
  Ear Infection-non-SAE, NR, Mild | 0.005 | 0.002
  Ear Infection-non-SAE, NR, Mod | 0.003 | 0.001
  Ear Pain-non-SAE, NR, Mild | 0.008 | 0.002
  Ear Pain-non-SAE, NR, Mod | 0 | 0.001
  Ecchymosis-non-SAE, NR, Mild | 0 | 0.001
  Eczema-non-SAE, NR, Mild | 0 | 0.001
  Eczema-non-SAE, NR, Mod | 0 | 0.001
  Eczema-non-SAE, NR, Severe | 0.003 | 0
  Eosinophil Count-non-SAE, NR, Mild | 0 | 0.001
  Epitaxis-non-SAE, NR, Mild | 0.005 | 0.003
  Epitaxis-non-SAE, NR, Mod | 0.005 | 0.002
  Erythema-non-SAE, NR, Mild | 0.003 | 0
  Erythema-non-SAE, RIGIV, Mod | 0 | 0.001
  Erythema-non-SAE, RrHu, Mild | 0 | 0.001
  Erythema-non-SAE, Rboth, Mild | 0 | 0.001
  Erythema-non-SAE, Rboth, Mod | 0 | 0.001
  Eustachian Tube Dysfunction-non-SAE, NR, Mild | 0.003 | 0
  Excoriation-non-SAE, NR, Mild | 0.005 | 0.002
  Extravasation Blood-non-SAE, Rboth, Mild | 0 | 0.001
  Eye Irritation-non-SAE, NR, Mild | 0 | 0.001
  Eye Pruritus-non-SAE, NR, Mod | 0 | 0.001
  Eye Swelling-non-SAE, NR, Mod | 0 | 0.001
  Fall-non-SAE, NR, Mild | 0 | 0.001
  Fall-non-SAE, NR, Mod | 0 | 0.001
  Fatigue-non-SAE, NR, Mild | 0.003 | 0.004
  Fatigue-non-SAE, NR, Mod | 0.003 | 0.002
  Fatigue-non-SAE, RIGIV, Mild | 0.022 | 0.007
  Fatigue-non-SAE, RIGIV, Mod | 0 | 0.003
  Fatigue-non-SAE, Rboth, Mild | 0 | 0.003
  Feeling Abnormal-non-SAE, Rboth, Mod | 0 | 0.001
  Feeling Cold-non-SAE, RIGIV, Mild | 0.005 | 0
  Flatulence-non-SAE, NR, Mild | 0 | 0.001
  Flatulence-non-SAE, NR, Mod | 0 | 0.001
  Food Poisoning-non-SAE, NR, Mod | 0 | 0.001
  Free Haemoglobin Present-non-SAE, NR, Mild | 0.003 | 0.001
  Free Haemoglobin Present-non-SAE, NR, Severe | 0.003 | 0

55. Secondary Outcome: Rate of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to Study Drug, and Severity Per Infusion (G-M)
Description: as for outcome 52
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Number of AEs per infusion
  Gait Disturbance-non-SAE, NR, Mild | 0 | 0.001
  Gastroenteritis-non-SAE, NR, Mild | 0 | 0.003
  Gastroenteritis-non-SAE, NR, Mod | 0.005 | 0.002
  Gastroenteritis-non-SAE, RIGIV, Mild | 0.003 | 0
  Gastroenteritis-SAE, NR, Mod | 0 | 0.001
  Gastroenteritis Bacterial-non-SAE, NR, Mod | 0 | 0.001
  Gastroenteritis Viral-non-SAE, NR, Mild | 0.008 | 0.005
  Gastroenteritis Viral-non-SAE, NR, Mod | 0 | 0.004
  Gastroenteritis Viral-non-SAE, RIGIV, Mild | 0 | 0.001
  Gastrointestinal Haemorrhage-non-SAE, NR, Severe | 0 | 0.001
  Gastrooesophageal Reflux Disease-non-SAE, NR, Mild | 0.003 | 0.002
  Gastrooesophageal Reflux Disease-non-SAE, NR, Mod | 0.003 | 0
  Genital Herpes-non-SAE, NR, Mild | 0.003 | 0
  Genital Swelling-non-SAE, Rboth, Mod | 0 | 0.001
  Goitre-non-SAE, NR, Mild | 0.003 | 0
  Gout-non-SAE, NR, Mild | 0 | 0.001
  Grand Mal Convulsion-non-SAE, NR, Severe | 0.003 | 0
  Grand Mal Convulsion-SAE, NR, Severe | 0 | 0.001
  Gravitational Oedema-non-SAE, Rboth, Mod | 0 | 0.001
  Groin Pain-non-SAE, NR, Mild | 0 | 0.001
  Groin Pain-non-SAE, RIGIV, Mild | 0 | 0.001
  Groin Pain-non-SAE, RrHu, Mod | 0 | 0.001
  Haematoma-non-SAE, NR, Mild | 0.003 | 0.001
  Haematoma-non-SAE, NR, Mod | 0 | 0.001
  Haematuria-non-SAE, NR, Mild | 0 | 0.001
  Haemoglobin Abnormal-non-SAE, NR, Mild | 0 | 0.001
  Haemorrhoids-non-SAE, NR, Mild | 0 | 0.002
  Hand Fracture-non-SAE, NR, Mod | 0 | 0.001
  Headache-non-SAE, NR, Mild | 0.036 | 0.014
  Headache-non-SAE, NR, Mod | 0.003 | 0.003
  Headache-non-SAE, NR, Severe | 0.003 | 0
  Headache-non-SAE, RIGIV, Mild | 0.068 | 0.012
  Headache-non-SAE, RIGIV, Mod | 0.033 | 0.004
  Headache-non-SAE, RIGIV, Severe | 0.003 | 0
  Headache-non-SAE, Rboth, Mild | 0 | 0.008
  Headache-non-SAE, Rboth, Mod | 0 | 0.007
  Headache-SAE, NR, Severe | 0 | 0.001
  Hearing Impaired-non-SAE, NR, Mild | 0 | 0.001
  Heart Rate Increased-non-SAE, RIGIV, Mild | 0.011 | 0
  Heat Rash-non-SAE, NR, Mild | 0 | 0.001
  Heat Stroke-non-SAE, NR, Mod | 0 | 0.001
  Herpes Simplex Ophthalmic-non-SAE, NR, Mod | 0 | 0.001
  Herpes Zoster-non-SAE, NR, Mod | 0 | 0.001
  Hiatus Hernia-non-SAE, NR, Mod | 0 | 0.001
  Hot Flush-non-SAE, RIGIV, Mild | 0.003 | 0
  Hyperaesthesia-non-SAE, NR, Mild | 0 | 0.001
  Hypercholesterolaemia-non-SAE, NR, Mod | 0 | 0.001
  Hyperkeratosis-non-SAE, NR, Mild | 0 | 0.001
  Hypertension-non-SAE, NR, Mod | 0 | 0.004
  Hypertension-non-SAE, RIGIV, Mild | 0 | 0.002
  Hypertension-non-SAE, RIGIV, Mod | 0 | 0.001
  Hypertonia-non-SAE, NR, Mild | 0 | 0.001
  Hypothyroidism-non-SAE, NR, Mild | 0 | 0.001
  Idiopathic Urticaria-non-SAE, NR, Mod | 0.003 | 0
  Increased Upper Airway Secretion-non-SAE, NR, Mild | 0.005 | 0
  Infected Bites-non-SAE, NR, Mild | 0 | 0.002
  Infected Bites-non-SAE, NR, Mod | 0.003 | 0.001
  Infection-non-SAE, NR, Mod | 0 | 0.002
  Influenza-non-SAE, NR, Mild | 0.003 | 0.002
  Influenza-non-SAE, NR, Mod | 0.011 | 0.003
  Influenza Like Illness-non-SAE, NR, Mild | 0 | 0.001
  Infusion Related Reaction-non-SAE, RIGIV, Mild | 0 | 0.001
  Infusion Related Reaction-non-SAE, RIGIV, Mod | 0.003 | 0
  Infusion Related Reaction-non-SAE, Rboth, Mild | 0 | 0.001
  Infusion Related Reaction-non-SAE, Rboth, Mod | 0 | 0.001
  Infusion Site Discomfort-non-SAE, RIGIV, Mild | 0 | 0.005
  Infusion Site Discomfort-non-SAE, RrHu, Mod | 0 | 0.001
  Infusion Site Discomfort-non-SAE, Rboth, Mild | 0 | 0.013
  Infusion Site Discomfort-non-SAE, Rboth, Mod | 0 | 0.007
  Infusion Site Erythema-non-SAE, RIGIV, Mild | 0 | 0.001
  Infusion Site Erythema-non-SAE, RrHu, Mild | 0 | 0.002
  Infusion Site Erythema-non-SAE, Rboth, Mild | 0 | 0.018
  Infusion Site Erythema-non-SAE, Rboth, Mod | 0 | 0.004
  Infusion Site Extravasation-non-SAE, NR, Mild | 0.005 | 0
  Infusion Site Haematoma-non-SAE, RIGIV, Mild | 0 | 0.001
  Infusion Site Haemorrhage-non-SAE, Rboth, Mild | 0 | 0.001
  Infusion Site Hypersensitivity-non-SAE, NR, Severe | 0 | 0.001
  Infusion Site Hypersensitivity-non-SAE, Rboth, Mod | 0 | 0.001
  Infusion Site Mass-non-SAE, RIGIV, Mild | 0 | 0.001
  Infusion Site Mass-non-SAE, Rboth, Mild | 0 | 0.002
  Infusion Site Oedema-non-SAE, Rboth, Mild | 0 | 0.004
  Infusion Site Oedema-non-SAE, Rboth, Mod | 0 | 0.004
  Infusion Site Pain-non-SAE, NR, Mild | 0 | 0.002
  Infusion Site Pain-non-SAE, RIGIV, Mild | 0.003 | 0.011
  Infusion Site Pain-non-SAE, RIGIV, Mod | 0 | 0.005
  Infusion Site Pain-non-SAE, RrHu, Mild | 0 | 0.031
  Infusion Site Pain-non-SAE, RrHu, Mod | 0 | 0.001
  Infusion Site Pain-non-SAE, Rboth, Mild | 0 | 0.017
  Infusion Site Pain-non-SAE, Rboth, Mod | 0 | 0.014
  Infusion Site Pain-non-SAE, Rboth, Severe | 0 | 0.001
  Infusion Site Pruritus-non-SAE, RIGIV, Mild | 0 | 0.002
  Infusion Site Pruritus-non-SAE, RrHu, Mild | 0 | 0.004
  Infusion Site Pruritus-non-SAE, Rboth, Mild | 0 | 0.005
  Infusion Site Pruritus-non-SAE, Rboth, Mod | 0 | 0.004
  Infusion Site Reaction-non-SAE, Rboth, Mild | 0 | 0.001
  Infusion Site Reaction-non-SAE, Rboth, Mod | 0 | 0.002
  Infusion Site Swelling-non-SAE, RIGIV, Mild | 0 | 0.002
  Infusion Site Swelling-non-SAE, Rboth, Mild | 0 | 0.003
  Infusion Site Swelling-non-SAE, Rboth, Mod | 0 | 0.004
  Infusion Site Swelling-non-SAE, Rboth, Severe | 0 | 0.001
  Infusion Site Warmth-non-SAE, Rboth, Mild | 0 | 0.002
  Ingrowing Nail-non-SAE, NR, Mod | 0 | 0.001
  Injection Site Erythema-non-SAE, RIGIV, Mild | 0 | 0.001
  Injury-non-SAE, NR, Mild | 0.003 | 0
  Insomnia-non-SAE, NR, Mild | 0.003 | 0
  Intervertebral Disc Protrusion-non-SAE, NR, Mod | 0.003 | 0
  Irritable Bowel Syndrome-non-SAE, NR, Mild | 0 | 0.001
  Irritable Bowel Syndrome-non-SAE, NR, Mod | 0 | 0.002
  Joint Effusion-non-SAE, NR, Mild | 0 | 0.001
  Joint Effusion-non-SAE, NR, Mod | 0 | 0.001
  Joint Injury-non-SAE, NR, Mod | 0.003 | 0.001
  Joint Range of Motion Decreased-non-SAE, NR, Mod | 0 | 0.002
  Joint Sprain-non-SAE, NR, Mild | 0 | 0.001
  Joint Sprain-non-SAE, NR, Mod | 0 | 0.002
  Joint Swelling-non-SAE, NR, Mild | 0 | 0.001
  Jugular Vein Distension-non-SAE, NR, Mild | 0 | 0.001
  Lethargy-non-SAE, NR, Mild | 0 | 0.001
  Lethargy-non-SAE, RIGIV, Mod | 0.003 | 0
  Ligament Injury-non-SAE, NR, Mod | 0 | 0.001
  Ligament Sprain-non-SAE, NR, Mod | 0 | 0.001
  Limb Injury-non-SAE, NR, Mild | 0.003 | 0
  Lip Injury-non-SAE, NR, Mild | 0 | 0.001
  Lip Ulceration-non-SAE, NR, Mild | 0 | 0.001
  Local Swelling-non-SAE, RIGIV, Mild | 0 | 0.003
  Local Swelling-non-SAE, Rboth, Mild | 0 | 0.003
  Localised Infection-non-SAE, NR, Mild | 0 | 0.001
  Localised Oedema-non-SAE, RIGIV, Mild | 0 | 0.001
  Localised Oedema-non-SAE, Rboth, Mod | 0 | 0.001
  Lung Infection-non-SAE, NR, Mod | 0.003 | 0
  Lung Infection-non-SAE, NR, Severe | 0.003 | 0
  Lymph Gland Infection-non-SAE, NR, Mod | 0.003 | 0
  Lymph Node Pain-non-SAE, NR, Mild | 0.003 | 0
  Lymph Node Pain-non-SAE, NR, Mod | 0 | 0.001
  Lymph Node Palpable-non-SAE, NR, Mild | 0.003 | 0
  Lymphadenitis-non-SAE, NR, Mod | 0.003 | 0
  Lymphadenopathy-non-SAE, NR, Mild | 0.005 | 0.007
  Lymphangitis-non-SAE, NR, Mod | 0 | 0.001
  Lymphocyte Count Decreased-non-SAE, RIGIV, Mild | 0 | 0.001
  Lymphoedema-non-SAE, NR, Severe | 0.003 | 0
  Malaise-non-SAE, NR, Mild | 0 | 0.002
  Malaise-non-SAE, NR, Mod | 0 | 0.001
  Malaise-non-SAE, RIGIV, Mod | 0.003 | 0
  Malaise-non-SAE, RrHu, Mild | 0 | 0.001
  Malaise-non-SAE, RrHu, Mod | 0 | 0.001
  Memory Impairment-non-SAE, NR, Mod | 0 | 0.001
  Migraine-non-SAE, NR, Mild | 0.003 | 0.001
  Migraine-non-SAE, NR, Mod | 0 | 0.002
  Migraine-non-SAE, NR, Severe | 0.003 | 0
  Migraine-non-SAE, RIGIV, Mild | 0.003 | 0.001
  Migraine-non-SAE, RIGIV, Mod | 0.003 | 0.004
  Migraine-non-SAE, RIGIV, Severe | 0 | 0.001
  Migraine-non-SAE, Rboth, Mod | 0 | 0.001
  Molluscum Contagiosum-non-SAE, NR, Mild | 0.005 | 0
  Mouth Ulceration-non-SAE, NR, Mild | 0.003 | 0
  Multiple Sclerosis Relapse-non-SAE, NR, Mod | 0 | 0.001
  Muscle Fatigue-non-SAE, NR, Mild | 0 | 0.001
  Muscle Injury-non-SAE, NR, Mild | 0 | 0.002
  Muscle Spasms-non-SAE, NR, Mild | 0 | 0.001
  Muscle Spasms-non-SAE, RIGIV, Mild | 0.003 | 0
  Muscle Strain-non-SAE, NR, Mild | 0.003 | 0.001
  Muscle Strain-non-SAE, NR, Mod | 0 | 0.001
  Muscular Weakness-non-SAE, NR, Mild | 0.003 | 0
  Musculoskeletal Chest Pain-non-SAE, NR, Mild | 0 | 0.001
  Musculoskeletal Chest Pain-non-SAE, RIGIV, Mild | 0 | 0.001
  Musculoskeletal Pain-non-SAE, NR, Mild | 0.005 | 0
  Musculoskeletal Pain-non-SAE, NR, Mod | 0.003 | 0.001
  Musculoskeletal Stiffness-non-SAE, NR, Mild | 0.003 | 0.001
  Myalgia-non-SAE, NR, Mild | 0.008 | 0.004
  Myalgia-non-SAE, NR, Mod | 0.003 | 0.004
  Myalgia-non-SAE, NR, Severe | 0 | 0.001
  Myalgia-non-SAE, RIGIV, Mild | 0 | 0.005
  Myalgia-non-SAE, RIGIV, Mod | 0.003 | 0.001
  Myalgia-non-SAE, Rboth, Mild | 0 | 0.003

56. Secondary Outcome: Rate of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to Study Drug, and Severity Per Infusion (N-Z)
Description: Categories presented as Preferred term-Seriousness, Relatedness, Severity. The following codes are to be used: Seriousness: non-SAE-non-serious AE; SAE-serious AE Relationship: NR-not related to immune globulin (IGIV), 10% and recombinant human hyaluronidase (rHuPH20); ; RIGIV-related to IGIV, 10%; RrHu-related to rHuPH20; Rboth-related to both IGIV, 10% and rHuPH20 Severity: Mild; Mod (Moderate); Severe Preferred terms abbreviated: Resp.-Respiratory WBC - White blood cells
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Number of AEs per infusion
  Nasal Congestion-non-SAE, NR, Mild | 0.011 | 0.003
  Nasal Congestion-non-SAE, NR, Mod | 0 | 0.002
  Nasal Congestion-non-SAE, RIGIV, Mild | 0 | 0.003
  Nasal Discomfort-non-SAE, NR, Mild | 0 | 0.001
  Nasal Mucosal Discolouration-non-SAE, NR, Mild | 0 | 0.001
  Nasal Turbinate Hypertrophy-non-SAE, NR, Mild | 0 | 0.001
  Nasopharyngitis-non-SAE, NR, Mild | 0.011 | 0.007
  Nausea-non-SAE, NR, Mild | 0.008 | 0.015
  Nausea-non-SAE, NR, Mod | 0.005 | 0.003
  Nausea-non-SAE, RIGIV, Mild | 0.019 | 0.001
  Nausea-non-SAE, RIGIV, Mod | 0.003 | 0
  Nausea-non-SAE, Rboth, Mild | 0 | 0.004
  Neck Pain-non-SAE, NR, Mild | 0.003 | 0.001
  Night Sweats-non-SAE, NR, Mild | 0.003 | 0
  Night Sweats-non-SAE, NR, Mod | 0 | 0.001
  Nodule-non-SAE, Rboth, Mild | 0 | 0.002
  Oedema-non-SAE, RIGIV, Mild | 0 | 0.001
  Oedema Genital-non-SAE, Rboth, Severe | 0 | 0.001
  Oedema Peripheral-non-SAE, NR, Mild | 0 | 0.001
  Oedema Peripheral-non-SAE, NR, Mod | 0 | 0.001
  Oedema Peripheral-non-SAE, Rboth, Mod | 0 | 0.002
  Oesophagitis-non-SAE, NR, Mild | 0 | 0.001
  Onychomycosis-non-SAE, NR, Mild | 0 | 0.001
  Oral Candidiasis-non-SAE, NR, Mod | 0 | 0.001
  Oral Fungal Infection-non-SAE, NR, Mild | 0 | 0.001
  Oral Herpes-non-SAE, NR, Mild | 0.003 | 0.002
  Oral Herpes-non-SAE, NR, Mod | 0 | 0.001
  Oral Pain-non-SAE, NR, Mild | 0 | 0.001
  Oral Pain-non-SAE, RrHu, Severe | 0 | 0.001
  Oropharyngeal Pain-non-SAE, NR, Mild | 0.003 | 0.004
  Oropharyngeal Pain-non-SAE, NR, Mod | 0.005 | 0.001
  Osteoarthritis-non-SAE, NR, Mod | 0 | 0.001
  Osteopenia-non-SAE, NR, Mild | 0 | 0.001
  Osteopenia-non-SAE, NR, Mod | 0 | 0.001
  Osteoporosis-non-SAE, NR, Mild | 0 | 0.001
  Otitis Externa-non-SAE, NR, Mild | 0 | 0.001
  Otitis Externa-non-SAE, NR, Mod | 0 | 0.001
  Otitis Media-non-SAE, NR, Mod | 0.003 | 0.001
  Pain-non-SAE, NR, Mild | 0.003 | 0.004
  Pain-non-SAE, NR, Mod | 0.003 | 0.001
  Pain-non-SAE, RIGIV, Mild | 0 | 0.001
  Pain-non-SAE, RIGIV, Mod | 0.005 | 0.001
  Pain-non-SAE, Rboth, Mild | 0 | 0.001
  Pain-non-SAE, Rboth, Mod | 0 | 0.001
  Pain in Extremity-non-SAE, NR, Mild | 0.005 | 0.001
  Pain in Extremity-non-SAE, NR, Mod | 0.003 | 0.002
  Pain in Extremity-non-SAE, RIGIV, Mod | 0.005 | 0
  Pain in Extremity-non-SAE, RIGIV, Severe | 0.003 | 0
  Pain in Extremity-non-SAE, Rboth, Mild | 0 | 0.003
  Pain in Extremity-non-SAE, Rboth, Mod | 0 | 0.002
  Palpitations-non-SAE, NR, Mild | 0.003 | 0.001
  Papule-non-SAE, NR, Mild | 0 | 0.001
  Peptic Ulcer Haemorrhage-SAE, NR, Severe | 0.003 | 0
  Periorbital Haematoma-non-SAE, NR, Mild | 0 | 0.001
  Peripheral Nerve Injury-non-SAE, NR, Mild | 0 | 0.001
  Pertussis-non-SAE, NR, Mod | 0 | 0.001
  Petit Mal Epilepsy-SAE, NR, Severe | 0 | 0.001
  Pharyngeal Erythema-non-SAE, NR, Mild | 0.003 | 0.003
  Pharyngitis-non-SAE, NR, Mild | 0.003 | 0.004
  Pharyngitis-non-SAE, NR, Mod | 0.003 | 0
  Pharyngitis Streptococcal-non-SAE, NR, Mod | 0 | 0.004
  Pneumonia-non-SAE, NR, Mild | 0 | 0.001
  Pneumonia-non-SAE, NR, Mod | 0 | 0.001
  Pneumonia Bacterial-non-SAE, NR, Mod | 0 | 0.001
  Post Procedural Infection-non-SAE, NR, Mild | 0.003 | 0.002
  Post Procedural Infection-non-SAE, NR, Mod | 0 | 0.004
  Postictal Paralysis-non-SAE, NR, Mod | 0 | 0.001
  Postoperative Wound Infection-non-SAE, NR, Mod | 0 | 0.001
  Procedural Pain-non-SAE, NR, Mild | 0 | 0.002
  Procedural Pain-non-SAE, NR, Mod | 0 | 0.001
  Productive Cough-non-SAE, NR, Mild | 0.003 | 0.001
  Pruritus-non-SAE, NR, Mild | 0.003 | 0
  Pruritus-non-SAE, RIGIV, Mild | 0.003 | 0
  Pruritus-non-SAE, Rboth, Mild | 0 | 0.001
  Pruritus-non-SAE, Rboth, Mod | 0 | 0.001
  Pruritus Generalized-non-SAE, NR, Mild | 0.003 | 0
  Pseudomonas Infection-non-SAE, NR, Mod | 0 | 0.001
  Psoriasis-non-SAE, NR, Mod | 0 | 0.001
  Pyrexia-non-SAE, NR, Mild | 0.008 | 0.010
  Pyrexia-non-SAE, NR, Mod | 0.005 | 0.001
  Pyrexia-non-SAE, RIGIV, Mild | 0.011 | 0.005
  Pyrexia-non-SAE, RIGIV, Mod | 0.005 | 0.002
  Pyrexia-non-SAE, Rboth, Mild | 0 | 0.002
  Rales-non-SAE, NR, Mild | 0 | 0.001
  Rales-non-SAE, NR, Mod | 0 | 0.001
  Rash-non-SAE, NR, Mild | 0.005 | 0.004
  Rash-non-SAE, NR, Mod | 0 | 0.001
  Rash Erythematous-non-SAE, NR, Mild | 0 | 0.001
  Rash Maculo-Papular-non-SAE, Rboth, Mild | 0 | 0.001
  Rash Pustular-non-SAE, NR, Mild | 0 | 0.001
  Rash Pustular-non-SAE, NR, Mod | 0.003 | 0
  Rash Papular-non-SAE, NR, Mild | 0 | 0.001
  Respiratory Failure-SAE, NR, Severe | 0 | 0.001
  Respiratory Rate Increased-non-SAE, NR, Mild | 0 | 0.001
  Respiratory Tract Congestion-non-SAE, NR, Mild | 0 | 0.001
  Respiratory Tract Infection-non-SAE, NR, Mild | 0.003 | 0.001
  Respiratory Tract Infection-non-SAE, NR, Mod | 0.003 | 0.003
  Respiratory Tract Infection Viral-non-SAE, NR, Mod | 0.003 | 0
  Rhinitis Allergic-non-SAE, NR, Mild | 0.003 | 0.003
  Rhinitis Allergic-non-SAE, NR, Mod | 0.008 | 0.001
  Rhinitis Allergic-non-SAE, RIGIV, Mod | 0.003 | 0
  Rhinorrhoea-non-SAE, NR, Mild | 0.003 | 0.001
  Road Traffic Accident-non-SAE, NR, Mod | 0 | 0.002
  Scleritis-non-SAE, NR, Mild | 0.003 | 0.001
  Scleritis-non-SAE, NR, Mod | 0 | 0.001
  Scratch-non-SAE, NR, Mild | 0.003 | 0
  Seborrhoeic Dermatitis-non-SAE, NR, Mild | 0 | 0.001
  Sicca Syndrome-non-SAE, NR, Mod | 0 | 0.001
  Sinus Congestion-non-SAE, NR, Mild | 0.003 | 0
  Sinus Headache-non-SAE, NR, Mild | 0.003 | 0
  Sinusitis-non-SAE, NR, Mild | 0.016 | 0.022
  Sinusitis-non-SAE, NR, Mod | 0.036 | 0.023
  Sinusitis-non-SAE, NR, Severe | 0 | 0.001
  Sinusitis-non-SAE, RIGIV, Mod | 0 | 0.001
  Skeletal Injury-non-SAE, NR, Mild | 0 | 0.001
  Skeletal Injury-non-SAE, NR, Mod | 0 | 0.001
  Skin Hyperpigmentation-non-SAE, Rboth, Mild | 0 | 0.001
  Skin Laceration-non-SAE, NR, Mild | 0 | 0.001
  Skin Laceration-non-SAE, NR, Mod | 0 | 0.001
  Skin Lesion-non-SAE, NR, Mild | 0.005 | 0.001
  Skin Lesion-non-SAE, NR, Mod | 0.003 | 0
  Skin Lesion-non-SAE, RIGIV, Mild | 0 | 0.002
  Skin Papilloma-non-SAE, NR, Mod | 0.003 | 0
  Spinal Osteoarthritis-non-SAE, NR, Mild | 0 | 0.002
  Squamous Cell Carcinoma-non-SAE, NR, Mod | 0.003 | 0.001
  Status Epilepticus-SAE, NR, Severe | 0 | 0.001
  Suicidal Ideation-non-SAE, NR, Mild | 0.003 | 0
  Sunburn-non-SAE, NR, Mild | 0 | 0.001
  Swelling-non-SAE, Rboth, Mild | 0 | 0.001
  Swelling-non-SAE, Rboth, Mod | 0 | 0.003
  Syncope-non-SAE, NR, Mild | 0 | 0.001
  Tachycardia-non-SAE, NR, Mild | 0 | 0.003
  Tachycardia-non-SAE, NR, Mod | 0 | 0.001
  Therapy Cessation-non-SAE, NR, Severe | 0 | 0.001
  Thrombosis-non-SAE, NR, Severe | 0 | 0.001
  Thrombosis-SAE, NR, Mod | 0 | 0.001
  Tinea Infection-non-SAE, NR, Mild | 0.005 | 0
  Tongue Coated-non-SAE, NR, Mild | 0 | 0.001
  Tonsillar Hypertrophy-non-SAE, NR, Mod | 0 | 0.001
  Tonsillar Hypertrophy-SAE, NR, Mild | 0 | 0.001
  Tooth Abscess-non-SAE, NR, Mild | 0.003 | 0
  Tooth Abscess-non-SAE, NR, Mod | 0 | 0.001
  Tooth Impacted-non-SAE, NR, Mod | 0 | 0.001
  Tooth Infection-non-SAE, NR, Mod | 0 | 0.001
  Toothache-non-SAE, NR, Mod | 0 | 0.001
  Tongue Injury-non-SAE, NR, Mild | 0 | 0.001
  Tremor-non-SAE, NR, Mild | 0 | 0.001
  Tricuspid Valve Incompetence-non-SAE, NR, Mild | 0 | 0.001
  Tympanic Membrane Disorder-non-SAE, NR, Mild | 0.003 | 0
  Tympanic Membrane Hyperaemia-non-SAE, NR, Mild | 0 | 0.002
  Upper Airway Cough Syndrome-non-SAE, NR, Mild | 0 | 0.001
  Upper Resp. Tract Infection-non-SAE, NR, Mild | 0.019 | 0.030
  Upper Resp. Tract Infection-non-SAE, NR, Mod | 0.005 | 0.009
  Urinary Tract Infection-non-SAE, NR, Mild | 0.003 | 0.002
  Urinary Tract Infection-non-SAE, NR, Mod | 0.014 | 0.004
  Urine Analysis Abnormal-non-SAE, NR, Mild | 0 | 0.001
  Urticaria-non-SAE, NR, Mild | 0 | 0.004
  Urticaria-non-SAE, NR, Mod | 0 | 0.001
  Urticaria-non-SAE, RIGIV, Mild | 0.003 | 0
  Uterine Polyp-non-SAE, NR, Mod | 0 | 0.001
  Vaginal Haemorrhage-non-SAE, NR, Mod | 0 | 0.001
  Vascular Access Complication-non-SAE, NR, Mild | 0.003 | 0
  Vertigo-non-SAE, NR, Mod | 0 | 0.001
  Viral Diarrhoea-non-SAE, NR, Mild | 0 | 0.001
  Viral Infection-non-SAE, NR, Mild | 0008 | 0.006
  Viral Infection-non-SAE, NR, Mod | 0.008 | 0.003
  Viral Infection-SAE, NR, Mild | 0.003 | 0
  Viral Upper Resp. Tract Infection-non-SAE, NR Mild | 0.003 | 0.007
  Viral Upper Resp. Tract Infection-non-SAE, NR, Mod | 0.003 | 0.001
  Vision Blurred-non-SAE, NR, Mild | 0 | 0.001
  Vitamin D Deficiency-non-SAE, NR, Mild | 0.003 | 0
  Vitamin D Deficiency-non-SAE, NR, Mod | 0 | 0.002
  Vomiting-non-SAE, NR, Mild | 0.014 | 0.006
  Vomiting-non-SAE, NR, Mod | 0 | 0.003
  Vomiting-non-SAE, RIGIV, Mild | 0.011 | 0.003
  Vomiting-non-SAE, RIGIV, Mod | 0.003 | 0.004
  Vomiting-non-SAE, RIGIV, Severe | 0.003 | 0
  Vomiting-non-SAE, Rboth, Mod | 0 | 0.001
  Vulvovaginal Pruritus-non-SAE, RIGIV, Mild | 0 | 0.001
  Weight Decreased-non-SAE, RrHu, Mild | 0 | 0.001
  Weight Decreased-non-SAE, RrHu, Mod | 0 | 0.001
  Wheezing-non-SAE, NR, Mod | 0 | 0.001
  WBC Count Decreased-non-SAE, RIGIV, Mild | 0 | 0.001
  White Blood Cells Urine Positive-non-SAE, NR, Mild | 0 | 0.001
  WBC Urine Positive-non-SAE, RIGIV Mild | 0.003 | 0

57. Secondary Outcome: Rate of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to Study Drug, and Severity Per Participant (A-F)
Description: as for outcome 51
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per participant
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number of AEs per participant
  Abdominal Discomfort-non-SAE, NR, Mod | 0 | 0.012
  Abdominal Distension-non-SAE, Rboth, Mild | 0 | 0.012
  Abdominal Hernia-non-SAE, NR, Mild | 0 | 0.012
  Abdominal Pain-non-SAE, NR, Mild | 0.011 | 0.025
  Abdominal Pain-non-SAE, NR, Mod | 0 | 0.012
  Abdominal Pain-non-SAE, Rboth, Mild | 0 | 0.037
  Abdominal Pain-non-SAE, Rboth, Mod | 0 | 0.012
  Abdominal Pain Lower-non-SAE, NR, Mild | 0 | 0.012
  Abdominal Pain Upper-non-SAE, NR, Mild | 0.011 | 0.062
  Abdominal Pain Upper-non-SAE, NR, Mod | 0.011 | 0
  Abdominal Pain Upper-non-SAE, RIGIV, Mild | 0 | 0.012
  Abdominal Pain Upper-non-SAE, RIGIV, Mod | 0.011 | 0
  Abdominal Pain Upper-non-SAE, Rboth, Mild | 0 | 0.025
  Abdominal Tenderness-non-SAE, NR, Mod | 0.011 | 0
  Abdominal Tenderness-non-SAE, RIGIV, Mild | 0 | 0.012
  Abdominal Tenderness-non-SAE, RIGIV, Mod | 0 | 0.025
  Acarodermatitis-non-SAE, NR, Mild | 0 | 0.012
  Acne-non-SAE, NR, Mild | 0.011 | 0.012
  Acute Sinusitis-non-SAE, NR, Mild | 0.011 | 0
  Acute Sinusitis-non-SAE, NR, Mod | 0 | 0.049
  Adenoidal Hypertrophy-non-SAE, NR, Mod | 0 | 0.012
  Adnexa Uteri Cyst-non-SAE, NR, Mild | 0.011 | 0
  Adrenocortical Insufficiency Acute-SAE, NR, Mod | 0 | 0.012
  Allergic Respiratory Symptom-non-SAE, NR, Mild | 0 | 0.012
  Allergic Sinusitis-non-SAE, NR, Mild | 0.011 | 0
  Alopecia-non-SAE, NR, Mild | 0.011 | 0
  Animal Bite-non-SAE, NR, Mod | 0.011 | 0
  Antibody Test Positive-non-SAE, Rboth, Mod | 0 | 0.012
  Anxiety-non-SAE, NR, Mild | 0 | 0.012
  Anxiety-non-SAE, NR, Mod | 0.011 | 0
  Aphthous Stomatitis-non-SAE, NR, Mild | 0.023 | 0.012
  Aphthous Stomatitis-non-SAE, NR, Mod | 0 | 0.012
  Arteriosclerosis Coronary Artery-non-SAE, NR, Mild | 0 | 0.012
  Arthralgia-non-SAE, NR, Mild | 0 | 0.062
  Arthralgia-non-SAE, NR, Mod | 0.011 | 0.074
  Arthralgia-non-SAE, RIGIV, Mild | 0 | 0.012
  Arthralgia-non-SAE, RIGIV, Mod | 0 | 0.025
  Arthritis-non-SAE, NR, Mod | 0.011 | 0.012
  Arthropathy-non-SAE, NR, Mod | 0.011 | 0
  Arthropod Bite-non-SAE, NR, Mild | 0.023 | 0.025
  Arthropod Sting-non-SAE, NR, Mild | 0 | 0.012
  Arthropod Sting-non-SAE, NR, Mod | 0.011 | 0
  Aspiration-non-SAE, NR, Mild | 0 | 0.012
  Asthenia-non-SAE, NR, Mild | 0 | 0.037
  Asthenia-non-SAE, NR, Mod | 0.011 | 0
  Asthenia-non-SAE, RIGIV, Mild | 0 | 0.012
  Asthma-non-SAE, NR, Mild | 0 | 0.049
  Asthma-non-SAE, NR, Mod | 0.092 | 0.259
  Asthma-non-SAE, NR, Severe | 0 | 0.012
  ADHD-non-SAE, NR, Mod | 0 | 0.012
  Back Injury-non-SAE, NR, Mod | 0.011 | 0
  Back Injury-SAE, NR, Severe | 0 | 0.012
  Back Pain-non-SAE, NR, Mild | 0.011 | 0.025
  Back Pain-non-SAE, NR, Mod | 0.011 | 0.062
  Bacterial Prostatitis-non-SAE, NR, Mild | 0 | 0.012
  Blepharitis-non-SAE, NR, Mod | 0.011 | 0
  Blister-non-SAE, NR, Mild | 0 | 0.012
  Blood Pressure Decreased-non-SAE, NR, Mild | 0 | 0.012
  Blood Pressure Decreased-non-SAE, Rboth, Mild | 0 | 0.012
  Blood Pressure Increased-non-SAE, NR, Mod | 0 | 0.012
  Blood Pressure Increased-non-SAE, RIGIV, Mild | 0 | 0.012
  Blood Pressure Increased-non-SAE, RIGIV, Mod | 0 | 0.012
  Blood Pressure Increased-non-SAE, RrHu, Mild | 0 | 0.012
  BP Systolic Increased-non-SAE, RIGIV, Mild | 0.011 | 0
  Blood Urea Increased-non-SAE, NR, Mild | 0 | 0.012
  Body Fat Disorder-non-SAE, NR, Mild | 0 | 0.012
  Body Tinea-non-SAE, NR, Mild | 0.011 | 0
  Body Tinea-non-SAE, NR, Mod | 0 | 0.012
  Bone Pain-non-SAE, NR, Mild | 0 | 0.012
  Breast Pain-non-SAE, NR, Mild | 0.011 | 0
  Bronchal Hyperreactivity-non-SAE, NR, Mild | 0 | 0.012
  Bronchitis-non-SAE, NR, Mild | 0.046 | 0.025
  Bronchitis-non-SAE, NR, Mod | 0.023 | 0.099
  Bronchitis-SAE, NR, Mod | 0.011 | 0
  Bronchospasm-non-SAE, NR, Mod | 0 | 0.012
  Burn Infection-non-SAE, NR, Mild | 0 | 0.012
  Burning Sensation-non-SAE, RIGIV, Mild | 0 | 0.012
  Burning Sensation-non-SAE, RIGIV, Mod | 0 | 0.012
  Burning Sensation-non-SAE, RrHu, Mild | 0 | 0.012
  Bursitis-non-SAE, NR, Mild | 0.011 | 0
  Bursitis-non-SAE, NR, Mod | 0 | 0.012
  Candidiasis-non-SAE, NR, Mild | 0.011 | 0
  Candidiasis-non-SAE, NR, Mod | 0.011 | 0.012
  Cardiac Murmur-non-SAE, NR, Mild | 0 | 0.012
  Cellulitis-non-SAE, NR, Mild | 0 | 0.012
  Cellulitis-non-SAE, NR, Mod | 0 | 0.037
  Cellulitis-non-SAE, Rboth, Mod | 0 | 0.012
  Cerumen Impaction-non-SAE, NR, Mild | 0 | 0.025
  Cervical Dysplasia-SAE, NR, Mild | 0.011 | 0.012
  Cheilitis-non-SAE, NR, Mild | 0.023 | 0
  Chest Pain-non-SAE, NR, Mild | 0 | 0.025
  Chills-non-SAE, NR, Mild | 0 | 0.037
  Chills-non-SAE, RIGIV, Mild | 0.069 | 0.012
  Chills-non-SAE, RIGIV, Mod | 0.034 | 0
  Chills-non-SAE, Rboth, Mild | 0 | 0.012
  COPD-non-SAE, NR, Mod | 0 | 0.025
  COPD-non-SAE, NR, Severe | 0.011 | 0
  Chronic Sinusitis-non-SAE, NR, Mild | 0 | 0.049
  Chronic Sinusitis-non-SAE, NR, Mod | 0.011 | 0.012
  Concussion-non-SAE, NR, Mod | 0.011 | 0
  Confusional State-non-SAE, NR, Mod | 0 | 0.012
  Confusional State-non-SAE, RIGIV, Mild | 0.011 | 0
  Conjunctivitis-non-SAE, NR, Mild | 0.011 | 0.025
  Conjunctivitis Allergic-non-SAE, NR, Mild | 0.011 | 0
  Conjunctivitis Allergic-non-SAE, NR, Mod | 0.011 | 0
  Conjunctivitis Bacterial-non-SAE, NR, Mild | 0.011 | 0.012
  Conjunctivitis Bacterial-non-SAE, NR, Mod | 0 | 0.012
  Conjunctivitis Bacterial-non-SAE, NR, Severe | 0 | 0.012
  Constipation-non-SAE, NR, Mild | 0 | 0.037
  Contusion-non-SAE, NR, Mild | 0.011 | 0.062
  Contusion-non-SAE, NR, Mod | 0.011 | 0
  Contusion-non-SAE, RIGIV, Mod | 0 | 0.012
  Coombs Test Positive-non-SAE, RIGIV, Mild | 0 | 0.012
  Costochondritis-non-SAE, NR, Mod | 0 | 0.012
  Cough-non-SAE, NR, Mild | 0.034 | 0.074
  Cough-non-SAE, NR, Mod | 0 | 0.025
  Cough-non-SAE, RIGIV, Mild | 0.011 | 0
  Cushingoid-non-SAE, NR, Mild | 0 | 0.012
  Cystitis-non-SAE, NR, Mild | 0 | 0.012
  Deafness Neurosensory-non-SAE, NR, Mild | 0.011 | 0
  Decreased Appetite-non-SAE, NR, Mild | 0.011 | 0.012
  Decreased Appetite-non-SAE, RrHu, Mild | 0 | 0.012
  Decreased Appetite-non-SAE, Rboth, Mild | 0 | 0.025
  Dehydration-non-SAE, NR, Mod | 0 | 0.025
  Dental Caries-non-SAE, NR, Mild | 0 | 0.025
  Dental Caries-non-SAE, NR, Mod | 0 | 0.037
  Depressed Mood-non-SAE, NR, Mild | 0 | 0.012
  Depression-non-SAE, NR, Severe | 0 | 0.012
  Dermal Cyst-non-SAE, NR, Mild | 0 | 0.012
  Dermatitis-non-SAE, NR, Mild | 0 | 0.025
  Dermatitis-non-SAE, NR, Mod | 0.011 | 0
  Dermatitis Acneiform-non-SAE, NR, Mod | 0.011 | 0
  Dermatitis Contact-non-SAE, NR, Mild | 0 | 0.025
  Dermatitis Contact-non-SAE, NR, Mod | 0.023 | 0.025
  Dermatitis Infected-non-SAE, NR, Mild | 0 | 0.025
  Dermatitis Infected-non-SAE, NR, Mod | 0 | 0.012
  Dermatitis Infected-non-SAE, NR, Severe | 0 | 0.012
  Device Failure-non-SAE, NR, Mild | 0.023 | 0.012
  Device Failure-non-SAE, NR, Mod | 0 | 0.025
  Diarrhoea-non-SAE, NR, Mild | 0.034 | 0.074
  Diarrhoea-non-SAE, NR, Mod | 0.023 | 0.049
  Diarrhoea-non-SAE, RIGIV, Mild | 0.011 | 0.012
  Diarrhoea-non-SAE, RIGIV, Mod | 0.011 | 0
  Diarrhoea Haemorrhagic-non-SAE, NR, Mild | 0.011 | 0
  Diarrhoea Infectious-non-SAE, NR, Mild | 0 | 0.012
  Diastolic Dysfunction-non-SAE, NR, Mild | 0 | 0.012
  Disaccharide Metabolism Disorder-non-SAE, NR, Mild | 0 | 0.012
  Disturbance in Attention-non-SAE, NR, Mild | 0 | 0.025
  Diverticulitis-non-SAE, NR, Mod | 0.011 | 0
  Dizziness-non-SAE, NR, Mild | 0.023 | 0.086
  Dizziness-non-SAE, NR, Mod | 0 | 0.025
  Dizziness-non-SAE, RIGIV, Mild | 0 | 0.037
  Dizziness-non-SAE, RIGIV, Mod | 0.011 | 0
  Drug Eruption-non-SAE, NR, Mod | 0.011 | 0
  Dry Eye-non-SAE, NR, Mod | 0 | 0.012
  Dry Mouth-non-SAE, NR, Mild | 0 | 0.012
  Dry Skin-non-SAE, NR, Mild | 0 | 0.037
  Dysmenorrhoea-non-SAE, NR, Mild | 0 | 0.012
  Dyspepsia-non-SAE, NR, Mild | 0 | 0.025
  Dyspepsia-non-SAE, NR, Mod | 0 | 0.012
  Dyspepsia-non-SAE, RIGIV, Mild | 0.011 | 0
  Dysphagia-non-SAE, NR, Mild | 0 | 0.012
  Dysphagia-non-SAE, NR, Mod | 0 | 0.012
  Dyspnoea-non-SAE, NR, Mild | 0.011 | 0
  Dyspnoea-non-SAE, NR, Mod | 0.011 | 0
  Dyspnoea-non-SAE, RIGIV, Mild | 0.011 | 0
  Dysuria-non-SAE, NR, Mild | 0 | 0.025
  Ear Infection-non-SAE, NR, Mild | 0.023 | 0.025
  Ear Infection-non-SAE, NR, Mod | 0.011 | 0.012
  Ear Pain-non-SAE, NR, Mild | 0.034 | 0.025
  Ear Pain-non-SAE, NR, Mod | 0 | 0.012
  Ecchymosis-non-SAE, NR, Mild | 0 | 0.012
  Eczema-non-SAE, NR, Mild | 0 | 0.012
  Eczema-non-SAE, NR, Mod | 0 | 0.012
  Eczema-non-SAE, NR, Severe | 0.011 | 0
  Eosinophil Count-non-SAE, NR, Mild | 0 | 0.012
  Epitaxis-non-SAE, NR, Mild | 0.023 | 0.037
  Epitaxis-non-SAE, NR, Mod | 0.023 | 0.025
  Erythema-non-SAE, NR, Mild | 0.011 | 0
  Erythema-non-SAE, RIGIV, Mod | 0 | 0.012
  Erythema-non-SAE, RrHu, Mild | 0 | 0.012
  Erythema-non-SAE, Rboth, Mild | 0 | 0.012
  Erythema-non-SAE, Rboth, Mod | 0 | 0.012
  Eustachian Tube Dysfunction-non-SAE, NR, Mild | 0.011 | 0
  Excoriation-non-SAE, NR, Mild | 0.025 | 0.025
  Extravasation Blood-non-SAE, Rboth, Mild | 0 | 0.012
  Eye Irritation-non-SAE, NR, Mild | 0 | 0.012
  Eye Pruritus-non-SAE, NR, Mod | 0 | 0.012
  Eye Swelling-non-SAE, NR, Mod | 0 | 0.012
  Fall-non-SAE, NR, Mild | 0 | 0.012
  Fall-non-SAE, NR, Mod | 0 | 0.012
  Fatigue-non-SAE, NR, Mild | 0.011 | 0.062
  Fatigue-non-SAE, NR, Mod | 0.011 | 0.025
  Fatigue-non-SAE, RIGIV, Mild | 0.092 | 0.099
  Fatigue-non-SAE, RIGIV, Mod | 0 | 0.037
  Fatigue-non-SAE, Rboth, Mild | 0 | 0.037
  Feeling Abnormal-non-SAE, Rboth, Mod | 0 | 0.012
  Feeling Cold-non-SAE, RIGIV, Mild | 0.023 | 0
  Flatulence-non-SAE, NR, Mild | 0 | 0.012
  Flatulence-non-SAE, NR, Mod | 0 | 0.012
  Food Poisoning-non-SAE, NR, Mod | 0 | 0.012
  Free Haemoglobin Present-non-SAE, NR, Mild | 0.011 | 0.012
  Free Haemoglobin Present-non-SAE, NR, Severe | 0.011 | 0

58. Secondary Outcome: Rate of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to Study Drug, and Severity Per Participant (G-M)
Description: as for outcome 52
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per participant
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number of AEs per participant
  Gait Disturbance-non-SAE, NR, Mild | 0 | 0.012
  Gastroenteritis-non-SAE, NR, Mild | 0 | 0.037
  Gastroenteritis-non-SAE, NR, Mod | 0.023 | 0.025
  Gastroenteritis-non-SAE, RIGIV, Mild | 0.011 | 0
  Gastroenteritis-SAE, NR, Mod | 0 | 0.012
  Gastroenteritis Bacterial-non-SAE, NR, Mod | 0 | 0.012
  Gastroenteritis Viral-non-SAE, NR, Mild | 0.034 | 0.074
  Gastroenteritis Viral-non-SAE, NR, Mod | 0 | 0.062
  Gastroenteritis Viral-non-SAE, RIGIV, Mild | 0 | 0.012
  Gastrointestinal Haemorrhage-non-SAE, NR, Severe | 0 | 0.012
  Gastrooesophageal Reflux Disease-non-SAE, NR, Mild | 0.011 | 0.025
  Gastrooesophageal Reflux Disease-non-SAE, NR, Mod | 0.011 | 0
  Genital Herpes-non-SAE, NR, Mild | 0.011 | 0
  Genital Swelling-non-SAE, Rboth, Mod | 0 | 0.012
  Goitre-non-SAE, NR, Mild | 0.011 | 0
  Gout-non-SAE, NR, Mild | 0 | 0.012
  Grand Mal Convulsion-non-SAE, NR, Severe | 0.011 | 0
  Grand Mal Convulsion-SAE, NR, Severe | 0 | 0.012
  Gravitational Oedema-non-SAE, Rboth, Mod | 0 | 0.012
  Groin Pain-non-SAE, NR, Mild | 0 | 0.012
  Groin Pain-non-SAE, RIGIV, Mild | 0 | 0.012
  Groin Pain-non-SAE, RrHu, Mod | 0 | 0.012
  Haematoma-non-SAE, NR, Mild | 0.011 | 0.012
  Haematoma-non-SAE, NR, Mod | 0 | 0.012
  Haematuria-non-SAE, NR, Mild | 0 | 0.012
  Haemoglobin Abnormal-non-SAE, NR, Mild | 0 | 0.012
  Haemorrhoids-non-SAE, NR, Mild | 0 | 0.025
  Hand Fracture-non-SAE, NR, Mod | 0 | 0.012
  Headache-non-SAE, NR, Mild | 0.149 | 0.198
  Headache-non-SAE, NR, Mod | 0.011 | 0.037
  Headache-non-SAE, NR, Severe | 0.011 | 0
  Headache-non-SAE, RIGIV, Mild | 0.287 | 0.173
  Headache-non-SAE, RIGIV, Mod | 0.138 | 0.062
  Headache-non-SAE, RIGIV, Severe | 0.011 | 0
  Headache-non-SAE, Rboth, Mild | 0 | 0.011
  Headache-non-SAE, Rboth, Mod | 0 | 0.099
  Headache-SAE, NR, Severe | 0 | 0.012
  Hearing Impaired-non-SAE, NR, Mild | 0 | 0.012
  Heart Rate Increased-non-SAE, RIGIV, Mild | 0.046 | 0
  Heat Rash-non-SAE, NR, Mild | 0 | 0.012
  Heat Stroke-non-SAE, NR, Mod | 0 | 0.012
  Herpes Simplex Ophthalmic-non-SAE, NR, Mod | 0 | 0.012
  Herpes Zoster-non-SAE, NR, Mod | 0 | 0.012
  Hiatus Hernia-non-SAE, NR, Mod | 0 | 0.012
  Hot Flush-non-SAE, RIGIV, Mild | 0.011 | 0
  Hyperaesthesia-non-SAE, NR, Mild | 0 | 0.012
  Hypercholesterolaemia-non-SAE, NR, Mod | 0 | 0.012
  Hyperkeratosis-non-SAE, NR, Mild | 0 | 0.012
  Hypertension-non-SAE, NR, Mod | 0 | 0.049
  Hypertension-non-SAE, RIGIV, Mild | 0 | 0.025
  Hypertension-non-SAE, RIGIV, Mod | 0 | 0.012
  Hypertonia-non-SAE, NR, Mild | 0 | 0.012
  Hypothyroidism-non-SAE, NR, Mild | 0 | 0.012
  Idiopathic Urticaria-non-SAE, NR, Mod | 0.011 | 0
  Increased Upper Airway Secretion-non-SAE, NR, Mild | 0.023 | 0
  Infected Bites-non-SAE, NR, Mild | 0 | 0.025
  Infected Bites-non-SAE, NR, Mod | 0.011 | 0.012
  Infection-non-SAE, NR, Mod | 0 | 0.025
  Influenza-non-SAE, NR, Mild | 0.011 | 0.025
  Influenza-non-SAE, NR, Mod | 0.046 | 0.037
  Influenza Like Illness-non-SAE, NR, Mild | 0 | 0.012
  Infusion Related Reaction-non-SAE, RIGIV, Mild | 0 | 0.012
  Infusion Related Reaction-non-SAE, RIGIV, Mod | 0.011 | 0
  Infusion Related Reaction-non-SAE, Rboth, Mild | 0 | 0.012
  Infusion Related Reaction-non-SAE, Rboth, Mod | 0 | 0.012
  Infusion Site Discomfort-non-SAE, RIGIV, Mild | 0 | 0.074
  Infusion Site Discomfort-non-SAE, RrHu, Mod | 0 | 0.012
  Infusion Site Discomfort-non-SAE, Rboth, Mild | 0 | 0.185
  Infusion Site Discomfort-non-SAE, Rboth, Mod | 0 | 0.099
  Infusion Site Erythema-non-SAE, RIGIV, Mild | 0 | 0.012
  Infusion Site Erythema-non-SAE, RrHu, Mild | 0 | 0.025
  Infusion Site Erythema-non-SAE, Rboth, Mild | 0 | 0.247
  Infusion Site Erythema-non-SAE, Rboth, Mod | 0 | 0.062
  Infusion Site Extravasation-non-SAE, NR, Mild | 0.023 | 0
  Infusion Site Haematoma-non-SAE, RIGIV, Mild | 0 | 0.012
  Infusion Site Haemorrhage-non-SAE, Rboth, Mild | 0 | 0.012
  Infusion Site Hypersensitivity-non-SAE, NR, Severe | 0 | 0.012
  Infusion Site Hypersensitivity-non-SAE, Rboth, Mod | 0 | 0.012
  Infusion Site Mass-non-SAE, RIGIV, Mild | 0 | 0.012
  Infusion Site Mass-non-SAE, Rboth, Mild | 0 | 0.025
  Infusion Site Oedema-non-SAE, Rboth, Mild | 0 | 0.049
  Infusion Site Oedema-non-SAE, Rboth, Mod | 0 | 0.062
  Infusion Site Pain-non-SAE, NR, Mild | 0 | 0.025
  Infusion Site Pain-non-SAE, RIGIV, Mild | 0.011 | 0.148
  Infusion Site Pain-non-SAE, RIGIV, Mod | 0 | 0.074
  Infusion Site Pain-non-SAE, RrHu, Mild | 0 | 0.432
  Infusion Site Pain-non-SAE, RrHu, Mod | 0 | 0.012
  Infusion Site Pain-non-SAE, Rboth, Mild | 0 | 0.235
  Infusion Site Pain-non-SAE, Rboth, Mod | 0 | 0.198
  Infusion Site Pain-non-SAE, Rboth, Severe | 0 | 0.012
  Infusion Site Pruritus-non-SAE, RIGIV, Mild | 0 | 0.025
  Infusion Site Pruritus-non-SAE, RrHu, Mild | 0 | 0.062
  Infusion Site Pruritus-non-SAE, Rboth, Mild | 0 | 0.074
  Infusion Site Pruritus-non-SAE, Rboth, Mod | 0 | 0.049
  Infusion Site Reaction-non-SAE, Rboth, Mild | 0 | 0.012
  Infusion Site Reaction-non-SAE, Rboth, Mod | 0 | 0.025
  Infusion Site Swelling-non-SAE, RIGIV, Mild | 0 | 0.025
  Infusion Site Swelling-non-SAE, Rboth, Mild | 0 | 0.037
  Infusion Site Swelling-non-SAE, Rboth, Mod | 0 | 0.049
  Infusion Site Swelling-non-SAE, Rboth, Severe | 0 | 0.012
  Infusion Site Warmth-non-SAE, Rboth, Mild | 0 | 0.025
  Ingrowing Nail-non-SAE, NR, Mod | 0 | 0.012
  Injection Site Erythema-non-SAE, RIGIV, Mild | 0 | 0.012
  Injury-non-SAE, NR, Mild | 0.011 | 0
  Insomnia-non-SAE, NR, Mild | 0.011 | 0
  Intervertebral Disc Protrusion-non-SAE, NR, Mod | 0.011 | 0
  Irritable Bowel Syndrome-non-SAE, NR, Mild | 0 | 0.012
  Irritable Bowel Syndrome-non-SAE, NR, Mod | 0 | 0.025
  Joint Effusion-non-SAE, NR, Mild | 0 | 0.012
  Joint Effusion-non-SAE, NR, Mod | 0 | 0.012
  Joint Injury-non-SAE, NR, Mod | 0.011 | 0.012
  Joint Range of Motion Decreased-non-SAE, NR, Mod | 0 | 0.025
  Joint Sprain-non-SAE, NR, Mild | 0 | 0.012
  Joint Sprain-non-SAE, NR, Mod | 0 | 0.025
  Joint Swelling-non-SAE, NR, Mild | 0 | 0.012
  Jugular Vein Distension-non-SAE, NR, Mild | 0 | 0.012
  Lethargy-non-SAE, NR, Mild | 0 | 0.012
  Lethargy-non-SAE, RIGIV, Mod | 0 | 0.011
  Ligament Injury-non-SAE, NR, Mod | 0 | 0.012
  Ligament Sprain-non-SAE, NR, Mod | 0 | 0.012
  Limb Injury-non-SAE, NR, Mild | 0.011 | 0
  Lip Injury-non-SAE, NR, Mild | 0 | 0.012
  Lip Ulceration-non-SAE, NR, Mild | 0 | 0.012
  Local Swelling-non-SAE, RIGIV, Mild | 0 | 0.037
  Local Swelling-non-SAE, Rboth, Mild | 0 | 0.037
  Localised Infection-non-SAE, NR, Mild | 0 | 0.012
  Localised Oedema-non-SAE, RIGIV, Mild | 0 | 0.012
  Localised Oedema-non-SAE, Rboth, Mod | 0 | 0.012
  Lung Infection-non-SAE, NR, Mod | 0.011 | 0
  Lung Infection-non-SAE, NR, Severe | 0.011 | 0
  Lymph Gland Infection-non-SAE, NR, Mod | 0.011 | 0
  Lymph Node Pain-non-SAE, NR, Mild | 0.011 | 0
  Lymph Node Pain-non-SAE, NR, Mod | 0 | 0.012
  Lymph Node Palpable-non-SAE, NR, Mild | 0.011 | 0
  Lymphadenitis-non-SAE, NR, Mod | 0.011 | 0
  Lymphadenopathy-non-SAE, NR, Mild | 0.023 | 0.099
  Lymphangitis-non-SAE, NR, Mod | 0 | 0.012
  Lymphocyte Count Decreased-non-SAE, RIGIV, Mild | 0 | 0.012
  Lymphoedema-non-SAE, NR, Severe | 0.011 | 0
  Malaise-non-SAE, NR, Mild | 0 | 0.025
  Malaise-non-SAE, NR, Mod | 0 | 0.012
  Malaise-non-SAE, RIGIV, Mod | 0.011 | 0
  Malaise-non-SAE, RrHu, Mild | 0 | 0.012
  Malaise-non-SAE, RrHu, Mod | 0 | 0.012
  Memory Impairment-non-SAE, NR, Mod | 0 | 0.012
  Migraine-non-SAE, NR, Mild | 0.011 | 0.012
  Migraine-non-SAE, NR, Mod | 0 | 0.025
  Migraine-non-SAE, NR, Severe | 0.011 | 0
  Migraine-non-SAE, RIGIV, Mild | 0.011 | 0.012
  Migraine-non-SAE, RIGIV, Mod | 0.011 | 0.049
  Migraine-non-SAE, RIGIV, Severe | 0 | 0.012
  Migraine-non-SAE, Rboth, Mod | 0 | 0.012
  Molluscum Contagiosum-non-SAE, NR, Mild | 0.023 | 0
  Mouth Ulceration-non-SAE, NR, Mild | 0.011 | 0
  Multiple Sclerosis Relapse-non-SAE, NR, Mod | 0 | 0.012
  Muscle Fatigue-non-SAE, NR, Mild | 0 | 0.012
  Muscle Injury-non-SAE, NR, Mild | 0 | 0.025
  Muscle Spasms-non-SAE, NR, Mild | 0 | 0.012
  Muscle Spasms-non-SAE, RIGIV, Mild | 0.011 | 0
  Muscle Strain-non-SAE, NR, Mild | 0.011 | 0.012
  Muscle Strain-non-SAE, NR, Mod | 0 | 0.012
  Muscular Weakness-non-SAE, NR, Mild | 0.011 | 0
  Musculoskeletal Chest Pain-non-SAE, NR, Mild | 0 | 0.012
  Musculoskeletal Chest Pain-non-SAE, RIGIV, Mild | 0 | 0.012
  Musculoskeletal Pain-non-SAE, NR, Mild | 0.023 | 0
  Musculoskeletal Pain-non-SAE, NR, Mod | 0.011 | 0.012
  Musculoskeletal Stiffness-non-SAE, NR, Mild | 0.011 | 0.012
  Myalgia-non-SAE, NR, Mild | 0.034 | 0.062
  Myalgia-non-SAE, NR, Mod | 0.011 | 0.049
  Myalgia-non-SAE, NR, Severe | 0 | 0.012
  Myalgia-non-SAE, RIGIV, Mild | 0 | 0.074
  Myalgia-non-SAE, RIGIV, Mod | 0.011 | 0.012
  Myalgia-non-SAE, Rboth, Mild | 0 | 0.037

59. Secondary Outcome: Rate of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to Study Drug, and Severity Per Participant (N-Z)
Description: as for outcome 53
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per participant
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number of AEs per participant
  Nasal Congestion-non-SAE, NR, Mild | 0.046 | 0.037
  Nasal Congestion-non-SAE, NR, Mod | 0 | 0.025
  Nasal Congestion-non-SAE, RIGIV, Mild | 0 | 0.037
  Nasal Discomfort-non-SAE, NR, Mild | 0 | 0.012
  Nasal Mucosal Discolouration-non-SAE, NR, Mild | 0 | 0.012
  Nasal Turbinate Hypertrophy-non-SAE, NR, Mild | 0 | 0.012
  Nasopharyngitis-non-SAE, NR, Mild | 0.046 | 0.099
  Nausea-non-SAE, NR, Mild | 0.034 | 0.210
  Nausea-non-SAE, NR, Mod | 0.023 | 0.037
  Nausea-non-SAE, RIGIV, Mild | 0.080 | 0.012
  Nausea-non-SAE, RIGIV, Mod | 0.011 | 0
  Nausea-non-SAE, Rboth, Mild | 0 | 0.049
  Neck Pain-non-SAE, NR, Mild | 0.011 | 0.012
  Night Sweats-non-SAE, NR, Mild | 0.011 | 0
  Night Sweats-non-SAE, NR, Mod | 0 | 0.012
  Nodule-non-SAE, Rboth, Mild | 0 | 0.025
  Oedema-non-SAE, RIGIV, Mild | 0 | 0.012
  Oedema Genital-non-SAE, Rboth, Severe | 0 | 0.012
  Oedema Peripheral-non-SAE, NR, Mild | 0 | 0.012
  Oedema Peripheral-non-SAE, NR, Mod | 0 | 0.012
  Oedema Peripheral-non-SAE, Rboth, Mod | 0 | 0.025
  Oesophagitis-non-SAE, NR, Mild | 0 | 0.012
  Onychomycosis-non-SAE, NR, Mild | 0 | 0.012
  Oral Candidiasis-non-SAE, NR, Mod | 0 | 0.012
  Oral Fungal Infection-non-SAE, NR, Mild | 0 | 0.012
  Oral Herpes-non-SAE, NR, Mild | 0.011 | 0.025
  Oral Herpes-non-SAE, NR, Mod | 0 | 0.012
  Oral Pain-non-SAE, NR, Mild | 0 | 0.012
  Oral Pain-non-SAE, RrHu, Severe | 0 | 0.012
  Oropharyngeal Pain-non-SAE, NR, Mild | 0.011 | 0.049
  Oropharyngeal Pain-non-SAE, NR, Mod | 0.023 | 0.012
  Osteoarthritis-non-SAE, NR, Mod | 0 | 0.012
  Osteopenia-non-SAE, NR, Mild | 0 | 0.012
  Osteopenia-non-SAE, NR, Mod | 0 | 0.012
  Osteoporosis-non-SAE, NR, Mild | 0 | 0.012
  Otitis Externa-non-SAE, NR, Mild | 0 | 0.012
  Otitis Externa-non-SAE, NR, Mod | 0 | 0.012
  Otitis Media-non-SAE, NR, Mod | 0.011 | 0.012
  Pain-non-SAE, NR, Mild | 0.011 | 0.062
  Pain-non-SAE, NR, Mod | 0.011 | 0.012
  Pain-non-SAE, RIGIV, Mild | 0 | 0.012
  Pain-non-SAE, RIGIV, Mod | 0.023 | 0.012
  Pain-non-SAE, Rboth, Mild | 0 | 0.012
  Pain-non-SAE, Rboth, Mod | 0 | 0.012
  Pain in Extremity-non-SAE, NR, Mild | 0.023 | 0.012
  Pain in Extremity-non-SAE, NR, Mod | 0.011 | 0.025
  Pain in Extremity-non-SAE, RIGIV, Mod | 0.023 | 0
  Pain in Extremity-non-SAE, RIGIV, Severe | 0.011 | 0
  Pain in Extremity-non-SAE, Rboth, Mild | 0 | 0.037
  Pain in Extremity-non-SAE, Rboth, Mod | 0 | 0.025
  Palpitations-non-SAE, NR, Mild | 0.011 | 0.012
  Papule-non-SAE, NR, Mild | 0 | 0.012
  Peptic Ulcer Haemorrhage-SAE, NR, Severe | 0.011 | 0
  Periorbital Haematoma-non-SAE, NR, Mild | 0 | 0.012
  Peripheral Nerve Injury-non-SAE, NR, Mild | 0 | 0.012
  Pertussis-non-SAE, NR, Mod | 0 | 0.012
  Petit Mal Epilepsy-SAE, NR, Severe | 0 | 0.012
  Pharyngeal Erythema-non-SAE, NR, Mild | 0.011 | 0.037
  Pharyngitis-non-SAE, NR, Mild | 0.011 | 0.049
  Pharyngitis-non-SAE, NR, Mod | 0.011 | 0
  Pharyngitis Streptococcal-non-SAE, NR, Mod | 0 | 0.049
  Pneumonia-non-SAE, NR, Mild | 0 | 0.012
  Pneumonia-non-SAE, NR, Mod | 0 | 0.012
  Pneumonia Bacterial-non-SAE, NR, Mod | 0 | 0.012
  Post Procedural Infection-non-SAE, NR, Mild | 0.011 | 0.025
  Post Procedural Infection-non-SAE, NR, Mod | 0 | 0.062
  Postictal Paralysis-non-SAE, NR, Mod | 0 | 0.012
  Postoperative Wound Infection-non-SAE, NR, Mod | 0 | 0.012
  Procedural Pain-non-SAE, NR, Mild | 0 | 0.025
  Procedural Pain-non-SAE, NR, Mod | 0 | 0.012
  Productive Cough-non-SAE, NR, Mild | 0.011 | 0.012
  Pruritus-non-SAE, NR, Mild | 0.011 | 0
  Pruritus-non-SAE, RIGIV, Mild | 0.011 | 0
  Pruritus-non-SAE, Rboth, Mild | 0 | 0.012
  Pruritus-non-SAE, Rboth, Mod | 0 | 0.012
  Pruritus Generalized-non-SAE, NR, Mild | 0.011 | 0
  Pseudomonas Infection-non-SAE, NR, Mod | 0 | 0.012
  Psoriasis-non-SAE, NR, Mod | 0 | 0.012
  Pyrexia-non-SAE, NR, Mild | 0.034 | 0.136
  Pyrexia-non-SAE, NR, Mod | 0.023 | 0.012
  Pyrexia-non-SAE, RIGIV, Mild | 0.046 | 0.074
  Pyrexia-non-SAE, RIGIV, Mod | 0.023 | 0.025
  Pyrexia-non-SAE, Rboth, Mild | 0 | 0.025
  Rales-non-SAE, NR, Mild | 0 | 0.012
  Rales-non-SAE, NR, Mod | 0 | 0.012
  Rash-non-SAE, NR, Mild | 0.023 | 0.062
  Rash-non-SAE, NR, Mod | 0 | 0.012
  Rash Erythematous-non-SAE, NR, Mild | 0 | 0.012
  Rash Maculo-Papular-non-SAE, Rboth, Mild | 0 | 0.012
  Rash Pustular-non-SAE, NR, Mild | 0 | 0.012
  Rash Pustular-non-SAE, NR, Mod | 0.011 | 0
  Rash Papular-non-SAE, NR, Mild | 0 | 0.012
  Respiratory Failure-SAE, NR, Severe | 0 | 0.012
  Respiratory Rate Increased-non-SAE, NR, Mild | 0 | 0.012
  Respiratory Tract Congestion-non-SAE, NR, Mild | 0 | 0.012
  Respiratory Tract Infection-non-SAE, NR, Mild | 0.011 | 0.012
  Respiratory Tract Infection-non-SAE, NR, Mod | 0.011 | 0.037
  Respiratory Tract Infection Viral-non-SAE, NR, Mod | 0.011 | 0
  Rhinitis Allergic-non-SAE, NR, Mild | 0.011 | 0.037
  Rhinitis Allergic-non-SAE, NR, Mod | 0.034 | 0.012
  Rhinitis Allergic-non-SAE, RIGIV, Mod | 0.011 | 0
  Rhinorrhoea-non-SAE, NR, Mild | 0.011 | 0.012
  Road Traffic Accident-non-SAE, NR, Mod | 0 | 0.025
  Scleritis-non-SAE, NR, Mild | 0.011 | 0.012
  Scleritis-non-SAE, NR, Mod | 0 | 0.012
  Scratch-non-SAE, NR, Mild | 0.011 | 0
  Seborrhoeic Dermatitis-non-SAE, NR, Mild | 0 | 0.012
  Sicca Syndrome-non-SAE, NR, Mod | 0 | 0.012
  Sinus Congestion-non-SAE, NR, Mild | 0.011 | 0
  Sinus Headache-non-SAE, NR, Mild | 0.011 | 0
  Sinusitis-non-SAE, NR, Mild | 0.069 | 0.309
  Sinusitis-non-SAE, NR, Mod | 0.149 | 0.321
  Sinusitis-non-SAE, NR, Severe | 0 | 0.012
  Sinusitis-non-SAE, RIGIV, Mod | 0 | 0.012
  Skeletal Injury-non-SAE, NR, Mild | 0 | 0.012
  Skeletal Injury-non-SAE, NR, Mod | 0 | 0.012
  Skin Hyperpigmentation-non-SAE, Rboth, Mild | 0 | 0.012
  Skin Laceration-non-SAE, NR, Mild | 0 | 0.012
  Skin Laceration-non-SAE, NR, Mod | 0 | 0.012
  Skin Lesion-non-SAE, NR, Mild | 0.023 | 0.012
  Skin Lesion-non-SAE, NR, Mod | 0.011 | 0
  Skin Lesion-non-SAE, RIGIV, Mild | 0 | 0.025
  Skin Papilloma-non-SAE, NR, Mod | 0.011 | 0
  Spinal Osteoarthritis-non-SAE, NR, Mild | 0 | 0.025
  Squamous Cell Carcinoma-non-SAE, NR, Mod | 0.011 | 0.012
  Status Epilepticus-SAE, NR, Severe | 0 | 0.012
  Suicidal Ideation-non-SAE, NR, Mild | 0.011 | 0
  Sunburn-non-SAE, NR, Mild | 0 | 0.012
  Swelling-non-SAE, Rboth, Mild | 0 | 0.012
  Swelling-non-SAE, Rboth, Mod | 0 | 0.037
  Syncope-non-SAE, NR, Mild | 0 | 0.012
  Tachycardia-non-SAE, NR, Mild | 0.037 | 0
  Tachycardia-non-SAE, NR, Mod | 0 | 0.012
  Therapy Cessation-non-SAE, NR, Severe | 0 | 0.012
  Thrombosis-non-SAE, NR, Severe | 0 | 0.012
  Thrombosis-SAE, NR, Mod | 0 | 0.012
  Tinea Infection-non-SAE, NR, Mild | 0 | 0.023
  Tongue Coated-non-SAE, NR, Mild | 0 | 0.012
  Tonsillar Hypertrophy-non-SAE, NR, Mod | 0 | 0.012
  Tonsillar Hypertrophy-SAE, NR, Mild | 0 | 0.012
  Tooth Abscess-non-SAE, NR, Mild | 0.011 | 0
  Tooth Abscess-non-SAE, NR, Mod | 0 | 0.012
  Tooth Impacted-non-SAE, NR, Mod | 0 | 0.012
  Tooth Infection-non-SAE, NR, Mod | 0 | 0.012
  Toothache-non-SAE, NR, Mod | 0 | 0.012
  Tongue Injury-non-SAE, NR, Mild | 0 | 0.012
  Tremor-non-SAE, NR, Mild | 0 | 0.012
  Tricuspid Valve Incompetence-non-SAE, NR, Mild | 0 | 0.012
  Tympanic Membrane Disorder-non-SAE, NR, Mild | 0.011 | 0
  Tympanic Membrane Hyperaemia-non-SAE, NR, Mild | 0 | 0.025
  Upper Airway Cough Syndrome-non-SAE, NR, Mild | 0 | 0.012
  Upper Resp. Tract Infection-non-SAE, NR, Mild | 0.080 | 0.420
  Upper Resp. Tract Infection-non-SAE, NR, Mod | 0.023 | 0.123
  Urinary Tract Infection-non-SAE, NR, Mild | 0.011 | 0.025
  Urinary Tract Infection-non-SAE, NR, Mod | 0.057 | 0.049
  Urine Analysis Abnormal-non-SAE, NR, Mild | 0 | 0.012
  Urticaria-non-SAE, NR, Mild | 0 | 0.062
  Urticaria-non-SAE, NR, Mod | 0 | 0.012
  Urticaria-non-SAE, RIGIV, Mild | 0.011 | 0
  Uterine Polyp-non-SAE, NR, Mod | 0 | 0.012
  Vaginal Haemorrhage-non-SAE, NR, Mod | 0 | 0.012
  Vascular Access Complication-non-SAE, NR, Mild | 0.011 | 0
  Vertigo-non-SAE, NR, Mod | 0 | 0.012
  Viral Diarrhoea-non-SAE, NR, Mild | 0 | 0.012
  Viral Infection-non-SAE, NR, Mild | 0.034 | 0.086
  Viral Infection-non-SAE, NR, Mod | 0.034 | 0.037
  Viral Infection-SAE, NR, Mild | 0.011 | 0
  Viral Upper Resp. Tract Infection-non-SAE, NR Mild | 0.011 | 0.099
  Viral Upper Resp. Tract Infection-non-SAE, NR, Mod | 0.011 | 0.012
  Vision Blurred-non-SAE, NR, Mild | 0 | 0.012
  Vitamin D Deficiency-non-SAE, NR, Mild | 0.011 | 0
  Vitamin D Deficiency-non-SAE, NR, Mod | 0 | 0.025
  Vomiting-non-SAE, NR, Mild | 0.057 | 0.096
  Vomiting-non-SAE, NR, Mod | 0 | 0.037
  Vomiting-non-SAE, RIGIV, Mild | 0.046 | 0.037
  Vomiting-non-SAE, RIGIV, Mod | 0.011 | 0.049
  Vomiting-non-SAE, RIGIV, Severe | 0.011 | 0
  Vomiting-non-SAE, Rboth, Mod | 0 | 0.012
  Vulvovaginal Pruritus-non-SAE, RIGIV, Mild | 0 | 0.012
  Weight Decreased-non-SAE, RrHu, Mild | 0 | 0.012
  Weight Decreased-non-SAE, RrHu, Mod | 0 | 0.012
  Wheezing-non-SAE, NR, Mod | 0 | 0.012
  WBC Count Decreased-non-SAE, RIGIV, Mild | 0 | 0.012
  White Blood Cells Urine Positive-non-SAE, NR, Mild | 0 | 0.012
  WBC Urine Positive-non-SAE, RIGIV Mild | 0.011 | 0

60. Secondary Outcome: Percentage of Infusions Associated With ≥1 AE Related to Either or Both Study Drugs
Description: Percentage of Infusions Associated With ≥1 AE Related to immune globulin intravenous (IGIV), 10%, [administered via intravenous (IV) or subcutaneous (SC) route], recombinant human hyaluronidase (rHuPH20) or both. The percentage of affected infusions is calculated per subject and then summarized by the median of all subjects analysed.
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Median (95% Confidence Interval); unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 With Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Percentage of infusions
  Including infections | 0.0 [0.0 to 25.0] | 8.3 [6.3 to 20.8]
  Excluding infections | 0.0 [0.0 to 25.0] | 8.3 [6.3 to 20.8]

61. Secondary Outcome: Percentage of Infusions Tolerated With IV and SC Administration at Dose Used in Study Epoch 2 (SC/rHuPH20 Treatment)
Description: Epoch 2: subcutaneous (SC) administration of immune globulin intravenous (IGIV), 10% with recombinant human hyaluronidase (rHuPH20) after ramp-up. Dose used in Epoch 2 (after ramp-up) was 108% of dose used in intravenous (IV) administration of IGIV, 10%. The percentage of affected infusions is calculated per subject and then summarized by the median of all subjects analysed.
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Median (95% Confidence Interval); unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Percentage of infusions | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

62. Secondary Outcome: Median Rate of AEs Temporally Associated or Related to Study Drug Per Infusion
Description: Temporally associated defined as during infusion or within 72 hours of completion of infusion. Related defined as determined by investigator to be at least possibly related to study drug (immune globulin intravenous [IGIV], 10% or recombinant human hyaluronidase [rHuPH20]). Expressed as a percentage.
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Median (95% Confidence Interval); unit: Percentage of AE
Units Other Than Participants: Infusions
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10% With rHuPH20 After Ramp-up
Number analyzed (Participants) | 87 | 81
Number analyzed (Infusions) | 365 | 1129
Percentage of AE
  Including Infections | 0.25 [0.25 to 0.50] | 0.22 [0.13 to 0.31]
  Excluding Infections | 0.25 [0.20 to 0.50] | 0.18 [0.12 to 0.26]

63. Secondary Outcome: Number of Participants Who Developed Neutralizing Antibodies to Recombinant Human Hyaluronidase (rHuPH20)
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Number of participants
Arm/Group | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 87
Number of participants | 0

64. Secondary Outcome: Percentage of Participants Who Developed Neutralizing Antibodies to Recombinant Human Hyaluronidase (rHuPH20)
Time Frame: Throughout the study period (17 months)
Population: Safety Analysis Data Set
Measure: Number; unit: Percentage of participants
Arm/Group | SC Administration of IGIV, 10% With rHuPH20
Number analyzed (Participants) | 81
Percentage of participants | 0.0

65. Secondary Outcome: Number of Participants Who Experienced a Hemoglobin Drop of >2.0 g/dL, With Evidence of Hemolysis on Further Analysis
Description: Further analysis for incidences of potential hemolysis included direct Coombs' test, free hemoglobin, serum haptoglobin, LDH, urine hemosiderin and microscopic urinalysis
Time Frame: Throughout the study period (17 months)
Measure: Number; unit: Number of participants
Groups:
- Participants in Safety Data Analysis Set: Participants exposed to either or both study drugs
Arm/Group | Participants in Safety Data Analysis Set
Number analyzed (Participants) | 87
Number of participants | 0

66. Secondary Outcome: Percentage of Participants Who Experienced a Hemoglobin Drop of >2.0 g/dL, With Evidence of Hemolysis on Further Analysis
Description: as for outcome 65
Time Frame: Throughout the study period (17 months)
Measure: Number; unit: Percentage of participants
Arm/Group | Participants in Safety Data Analysis Set
Number analyzed (Participants) | 87
Percentage of participants | 0

ADVERSE EVENTS:
Groups:
- IV Administration of IGIV, 10%: Consists of Pharmacokinetics (PK) of Intravenous (IV) treatment and efficacy and tolerability of IV infusions of immune globulin intravenous (IGIV), 10%.
- SC Administration of IGIV, 10%, With rHuPH20 (With Ramp-up): Consists of participants treated SC with IGIV, 10% at 108% of IV dose during administration of IGIV, 10%. This arm INCLUDES participants during ramp-up. Ramp-up: Participants were treated with SC infusions of IGIV, 10% with recombinant human hyaluronidase (rHuPH20). Treatment intervals and doses used for initial infusions were gradually increased during first weeks of treatment to allow participants to adjust to increasing volume administered SC. During SC administration of IGIV, 10% with rHuPh20, aim was to treat participants SC at same intervals (ie, every 3 or 4 weeks) as treated IV.
Arm/Group | IV Administration of IGIV, 10% | SC Administration of IGIV, 10%, With rHuPH20 (With Ramp-up)
Serious Adverse Events (participants affected / at risk) | 3/87 | 12/83
Other Adverse Events (participants affected / at risk) | 67/87 | 81/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Administration of IGIV, 10% (N=87) | SC Administration of IGIV, 10%, With rHuPH20 (With Ramp-up) (N=83)
Adrenocortical Insufficiency Acute (Endocrine disorders) | 0 (0) | 1 (1)
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Grand Mal Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Petit Mal Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Status Epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Cervical Dysplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Leukoplakia Oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Localised Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Administration of IGIV, 10% (N=87) | SC Administration of IGIV, 10%, With rHuPH20 (With Ramp-up) (N=83)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2 (2) | 7 (9)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 7 (10)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (3) | 6 (11)
DIARRHOEA (Gastrointestinal disorders) | 7 (7) | 10 (15)
NAUSEA (Gastrointestinal disorders) | 12 (13) | 15 (28)
VOMITING (Gastrointestinal disorders) | 8 (11) | 13 (21)
CHILLS (General disorders) | 7 (9) | 2 (6)
FATIGUE (General disorders) | 8 (10) | 14 (25)
INFUSION SITE DISCOMFORT (General disorders) | 0 (0) | 10 (33)
INFUSION SITE ERYTHEMA (General disorders) | 0 (0) | 14 (47)
INFUSION SITE OEDEMA (General disorders) | 0 (0) | 6 (16)
INFUSION SITE PAIN (General disorders) | 1 (1) | 37 (129)
INFUSION SITE PRURITUS (General disorders) | 0 (0) | 6 (21)
INFUSION SITE SWELLING (General disorders) | 0 (0) | 6 (13)
LOCAL SWELLING (General disorders) | 0 (0) | 5 (6)
PAIN (General disorders) | 4 (4) | 7 (13)
PYREXIA (General disorders) | 8 (11) | 13 (26)
BRONCHITIS (Infections and infestations) | 6 (6) | 8 (12)
CELLULITIS (Infections and infestations) | 0 (0) | 5 (5)
CHRONIC SINUSITIS (Infections and infestations) | 1 (1) | 5 (6)
GASTROENTERITIS (Infections and infestations) | 3 (3) | 5 (5)
GASTROENTERITIS VIRAL (Infections and infestations) | 3 (3) | 9 (12)
INFLUENZA (Infections and infestations) | 5 (5) | 5 (6)
NASOPHARYNGITIS (Infections and infestations) | 4 (4) | 5 (10)
POST PROCEDURAL INFECTION (Infections and infestations) | 1 (1) | 7 (7)
SINUSITIS (Infections and infestations) | 14 (19) | 35 (59)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (9) | 32 (49)
URINARY TRACT INFECTION (Infections and infestations) | 6 (6) | 7 (7)
VIRAL INFECTION (Infections and infestations) | 3 (6) | 9 (10)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 7 (11)
CONTUSION (Injury, poisoning and procedural complications) | 2 (2) | 6 (8)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 13 (16)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (8)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (5) | 11 (21)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (9)
DIZZINESS (Nervous system disorders) | 3 (3) | 11 (14)
HEADACHE (Nervous system disorders) | 24 (53) | 27 (63)
MIGRAINE (Nervous system disorders) | 3 (4) | 6 (14)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 14 (28)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (8)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (10)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (7)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (6)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
HYPERTENSION (Vascular disorders) | 0 (0) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 12 months after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥30 days prior to submission or communication. Baxter may request an additional delay of ≤60 days eg, for intellectual property protection